219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# CLINICAL STUDY PROTOCOL SPONSOR:

GlaxoSmithKline Biologicals SA (GSK)

**Primary study intervention** GSK's mRNA Clinical Research CR-04

Other study intervention Placebo (normal saline)

Study identifier 219112 (MRNA CLINRES-001)

NCT identifier number NCT05972993

IND number 29606

**Date of protocol** Final: 11 May 2023

**Date of protocol amendment** Amendment 3 Final: 07 Feb 2024

**Title** Exploratory, FTIH, observer-blind, randomized,

controlled study to evaluate safety, reactogenicity and immunogenicity of various doses of GSK's investigational mRNA-CR-04 vaccine when

administered intramuscularly in healthy adults 18 to

49 years of age

**Brief title** A safety and immune response study to evaluate

varying doses of an mRNA vaccine against COVID-

19 in healthy adults

**Sponsor signatory** Pavitra Keshavan, Sr. Director, Clinical Project

Lead, Vaccines Clinical Sciences

Based on GSK Protocol WS v17.3

©2024 GSK group of companies or its licensor.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# PROTOCOL AMENDMENT 3 INVESTIGATOR AGREEMENT

## I agree:

- To conduct the study in compliance with this protocol, any future protocol amendments, or protocol administrative changes, with the terms of the clinical trial agreement and with any other study conduct procedures and/or study conduct documents provided by GSK and/or CRO.
- To assume responsibility for the proper conduct of the study at this site.
- That I am aware of, and will comply with, GCP and all applicable regulatory requirements.
- That I will comply with the terms of the site agreement.
- To comply with local bio-safety legislation.
- To ensure that all persons assisting me with the study are adequately informed about the GSK study intervention and other study-related duties and functions as described in the protocol.
- To supervise any individual or party to whom I have delegated study-related duties and functions conducted at the study site.
- To ensure that any individual or party to whom I have delegated study-related duties and functions conducted at the study site are qualified to perform those study-related duties and functions.
- To acquire the reference ranges for laboratory tests performed locally and, if required by local regulations, obtain the laboratory's current certification or Quality Assurance procedure manual.
- To ensure that no clinical samples (including serum samples) are retained onsite or elsewhere without the approval of GSK and the express written informed consent of the participant.
- To perform no biological assays on the clinical samples other than those described in the protocol or its amendment(s).
- To co-operate with representative(s) of GSK in the monitoring process of the study and in resolution of queries about the data.
- To have control of all essential documents and records generated under my responsibility before, during, and after the study.
- That I have been informed that certain regulatory authorities require the sponsor to obtain and supply, as necessary, details about the investigator(s)' ownership interest in the sponsor or the investigational intervention(s), and more generally about their financial ties with the sponsor. GSK will use and disclose the information solely for the purpose of complying with regulatory requirements.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# Hence, I:

- Agree to supply GSK with any necessary information regarding ownership interest and financial ties (including those of my spouse and dependent children).
- Agree to promptly update this information if any relevant changes occur during the study and for 1 year following completion of the study.
- Agree that GSK may disclose any information about such ownership interests and financial ties to regulatory authorities.
- Agree to provide GSK with an updated Curriculum Vitae and all other documents required by regulatory agencies for this study.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| | Protocol Amendment 3 Fina |
|---|---|
| eTrack study number and abbreviated title | 219112 (MRNA CLINRES-001) |
| NCT identifier number | NCT05972993 |
| IND number | 29606 |
| Date of protocol | Final: 11 May 2023 |
| Date of protocol amendment | Amendment 3 Final: 07 Feb 2024 |
| Title | Exploratory, FTIH, observer-blind, randomized, controlled study to evaluate safety, reactogenicity and immunogenicity of various doses of GSK's investigational mRNA-CR-04 vaccine when administered intramuscularly in healthy adults 18 to 49 years of age |
| Investigator name | |
| Signature | |

4

07 Feb 2024

Date

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# **SPONSOR INFORMATION**

# 1. Sponsor

GSK (Rixensart)

# 2. Sponsor medical expert for the study

Refer to the local study contact information document.

# 3. Sponsor study monitor

Refer to the local study contact information document.

# 4. Sponsor study contact for reporting of SAEs

Back up study contact for reporting SAEs: refer to Section 8.4.7.

Study contact for reporting SAEs: refer to the local study contact information document.

# 5. Emergency unblinding

Refer to Section 6.3.4.

07 Feb 2024

5

# PROTOCOL AMENDMENT 3 SUMMARY OF CHANGES TABLE

## DOCUMENT HISTORY

| Document | Date | Substantial | Region |
|-------------------|-------------|-------------|--------------------|
| Amendment 3 | 07 Feb 2024 | Yes | United States (US) |
| Amendment 2 | 15 Nov 2023 | Yes | United States (US) |
| Amendment 1 | 03 Oct 2023 | Yes | United States (US) |
| Original Protocol | 11 May 2023 | - | - |

## **Overall Rationale for the Amendment:**

The Protocol Amendment 3 has been amended to allow for additional Day 31 interim analyses and to add a Part B to the study following the Day 15 interim analysis, during which a lower dose (3  $\mu$ g) of the mRNA-CR-04 vaccine will be evaluated and sponsor personnel will be unblinded.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Section 1.1 (Synopsis), Section 1.2 (Schema), Section 4.1 (Overall design), Section 4.2 (Scientific rationale for study design), Section 4.3 (Justification for dose), and Section 6.3.3 (Intervention allocation to the participant). | This study is divided into two parts (Parts A and B). Part B will commence only after all Part A participants have completed their Day 15 study visits and the Day 15 interim analysis is completed. In Part B, 42 more participants will be enrolled in parallel and randomly assigned in a 3:3:1 ratio to receive: (a) 3 µg mRNA-CR-04 vaccine, or (b) 10 µg mRNA-CR-04 vaccine, or (c) saline placebo. | To explore a wider range of vaccine doses and to repeat the 10 µg dose vaccine group, which may assist in standardizing the Part B to Part A study groups. |
| Section 1.1 (Synopsis), Section 1.2 (Schema), Section 4.1 (Overall design), Section 6.3.4 (Blinding and unblinding), Section 8.3.7.1 (Staggered administration of study intervention), Section 8.3.7.4 (SRT and iSRC evaluation), and Section 8.4.4.2.1 (Myocarditis and pericarditis: definitions and assessment). | Text modified to allow unblinding of sponsor personnel (including the SRT) to individual level treatment assignments following the Part A Day 15 interim analysis. The observer-blind will be maintained at the site level. | Practical consideration to allow all sponsor personnel to use unblinded data analyses from this initial phase 1 trial to plan further clinical development of the investigational vaccine platform. The SRT will no longer need to rely on the iSRC as the sole reviewer of unblinded safety data. |
| Section 2.2 (Background) and Section 4.3 (Justification for dose). | FDA authorization of monovalent<br>COVID-19 vaccine boosters<br>encoding XBB.1.5 since 11<br>September 2023 added to text. | Since the prior protocol<br>amendment, the FDA has<br>approved and authorized new<br>monovalent COVID-19 vaccines<br>encoding this variant for<br>administration as booster doses. |
| Section 6.1 (Study interventions administered). | Added a new table to specify the study interventions to be administered to Part B study participants. | To align with the new interventions planned for Part B of the study. |
| Section 8.2.3 (Immunological readouts). | Revised the number of participants column to add the planned 42 Part B study participants. | To align with the planned additional study participants in Part B of the study. |
| Section 9.3 (Analysis sets). | Modified the per protocol analysis set definition to clarify the immunogenicity endpoint of interest | To align the per protocol set definition immunogenicity endpoint of interest with the endpoint |

# 219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| | being the neutralizing antibody titer against pseudovirus bearing S protein and removed the overall safety analysis set. | specified in the statistical analysis plan and to remove the redundant overall safety analysis set. |
| Section 9.4.1 (Primary endpoint),<br>Section 9.4.2.1 (Safety endpoints),<br>Section 9.4.2.2 (Immunogenicity<br>endpoints), and Section 9.4.3<br>(Analyses of exploratory<br>immunogenicity endpoints). | Clarified that these statistical analyses will be performed descriptively and separately for study Part A and Part B participants and will be pooled for model based analyses. | To align with the additional analyses required with the addition of the study Part B participants. |
| Section 9.5.1 (Sequence of analyses). | Added text to perform a Day 31 interim analysis on Part A participants and to allow for potential Day 15 and Day 31 interim analyses for Part B participants. | To explicitly note the known and potential additional interim analyses currently planned for this study. |
| Throughout | Minor editorial and document formatting revisions. | Minor, therefore not summarized. |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# **TABLE OF CONTENTS**

| PR | отос | OL AMENDMENT 3 INVESTIGATOR AGREEMENT | 2 |
|---|---|---|---|
| SP | ONSO | R INFORMATION | 5 |
| PR | отос | OL AMENDMENT 3 SUMMARY OF CHANGES TABLE | 6 |
| LIS | TOF | ABBREVIATIONS AND DEFINITION OF TERMS | 15 |
| 1. | PRO <sup>-</sup> | TOCOL SUMMARY | 24 |
| | 1.1. | Synopsis | |
| | 1.2. | Schema | |
| | 1.3. | Schedule of Activities (SoA) | |
| 2. | INTR | ODUCTION | 31 |
| | 2.1. | Study rationale | |
| | 2.2. | Background | |
| | 2.3. | Benefit/risk assessment | |
| 3. | OBJE | ECTIVES, ENDPOINTS, AND ESTIMANDS | 34 |
| 4. | STUE | DY DESIGN | 35 |
| | 4.1. | Overall design | |
| | 4.2. | Scientific rationale for study design | |
| | 4.3. | Justification for dose | |
| | 4.4. | End-of-study definition | 38 |
| 5. | STUE | DY POPULATION | 38 |
| | 5.1. | Inclusion criteria | 39 |
| | 5.2. | Exclusion criteria | 39 |
| | | 5.2.1. Medical conditions | 39 |
| | | 5.2.2. Prior/concomitant therapy | 41 |
| | | 5.2.3. Other exclusions | |
| | 5.3. | Screen failures | 41 |
| | 5.4. | Criteria for temporarily delaying enrollment, randomization and study intervention administration | 42 |
| 6. | STUE | OY INTERVENTION AND CONCOMITANT THERAPY | 42 |
| | 6.1. | Study interventions administered | 42 |
| | 6.2. | Preparation, handling, storage, and accountability | 45 |
| | 6.3. | Measures to minimize bias: randomization and blinding | |
| | | 6.3.1. Participant identification | |
| | | 6.3.2. Randomization to study intervention | 45 |
| | | 6.3.3. Intervention allocation to the participant | |
| | | 6.3.4. Blinding and unblinding | 45 |
| | 6.4. | Study intervention compliance | |
| | 6.5. | Dose modification | |
| | 6.6. | Continued access to study intervention after the end of the study | |
| | 6.7. | Treatment of overdose | |
| | 6.8. | Concomitant therapy | 47 |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| 7. | | | ATION OF STUDY INTERVENTION AND PARTICIPANT | 40 |
|---|---|---|---|---|
| | | | ATION/WITHDRAWAL | |
| | 7.1. | | tinuation of study intervention | 48 |
| | | 7.1.1. | - J | 4.0 |
| | | | administration | |
| | 7.2. | | oant discontinuation/withdrawal from the study | |
| | 7.3. | Lost to | follow-up | 49 |
| 0 | СТИГ | N/ ACCE( | COMENTS AND DECCEPTIBES | 40 |
| 8. | 8.1. | | SSMENTS AND PROCEDURES | |
| | 0.1. | 8.1.1. | strative procedures Collection of demographic data | |
| | | 8.1.1.<br>8.1.2. | | |
| | | 8.1.3. | , | 50 |
| | | 0.1.5. | devices | 50 |
| | 8.2. | Immun | ogenicity assessments | |
| | 0.2. | 8.2.1. | Biological samples | |
| | | 8.2.2. | Laboratory assays | |
| | | 8.2.3. | Immunological read-outs | |
| | | 8.2.4. | Cytology | |
| | | 8.2.5. | Immunological correlates of protection | |
| | 8.3. | | assessments | |
| | 0.0. | 8.3.1. | Physical examination | |
| | | 8.3.2. | Pre-dosing body temperature | |
| | | 8.3.3. | Pregnancy test | |
| | | 8.3.4. | EKGs | |
| | | 8.3.5. | Warnings and precautions to administration of study | |
| | | | intervention | 56 |
| | | 8.3.6. | Clinical safety laboratory tests | |
| | | 8.3.7. | Study holding rules and safety monitoring | 57 |
| | | | 8.3.7.1. Staggered administration of study intervention | 57 |
| | | | 8.3.7.2. Outcome of safety evaluation | |
| | | | 8.3.7.3. Study holding rules | |
| | | | 8.3.7.4. SRT and iSRC evaluation | |
| | | 8.3.8. | Cardiac adjudication | |
| | 8.4. | AEs, S | AEs, and other safety reporting | 63 |
| | | 8.4.1. | Time period and frequency for collecting AE, SAE and | |
| | | | other safety information | 63 |
| | | 8.4.2. | Method of detecting AEs and SAEs | |
| | | 8.4.3. | Follow-up of AEs and SAEs | |
| | | 8.4.4. | AESI | |
| | | | 8.4.4.1. pIMDs | |
| | | | 8.4.4.2. Other AESIs | / 1 |
| | | | 8.4.4.2.1. Myocarditis and pericarditis: | 7.4 |
| | | | definitions and assessment | 71 |
| | | | 8.4.4.2.2. SARS-CoV-2 infection and | |
| | | | COVID-19 definitions and | 70 |
| | | 0 1 5 | assessment | |
| | | 8.4.5. | Regulatory reporting requirements for SAEs/AESIs | |
| | | 8.4.6.<br>8.4.7. | Pregnancy | / 5 |
| | | 0.4.7. | Contact information for reporting SAEs, AESIs, | 76 |
| | | 8.4.8. | pregnancies and study holding rules<br>Participant card | |
| | | U. <del>T</del> .U. | i arnopalit varu | |

| 219112 | (MRNA CLINRES-001) | ١ |
|--------|-----------------------|---|
| Proto | col Amendment 3 Final | ĺ |

| | | | 1 Totocol Amendment | o i iiiai |
|---|---|---|---|---|
| | 8.5. | | cokinetics | |
| | 8.6. | | S | |
| | 8.7. | | ers | |
| | 8.8. | | genicity assessments | |
| | 8.9. | | outcomes | |
| | 8.10. | Study pr | ocedures during special circumstances | / / |
| 9. | STATI | STICAL ( | CONSIDERATIONS | 78 |
| | 9.1. | Statistica | al hypotheses | 78 |
| | 9.2. | Sample | size determination | 78 |
| | 9.3. | Analysis | sets | |
| | | 9.3.1. | Criteria for elimination from analysis | |
| | 9.4. | | al analyses | |
| | | 9.4.1. | Primary endpoint | |
| | | 9.4.2. | Secondary endpoints/estimands analyses | |
| | | | 9.4.2.1. Safety endpoints | |
| | | | 9.4.2.2. Immunogenicity endpoints | |
| | | 9.4.3. | Analyses of exploratory immunogenicity endpoints | |
| | 9.5. | | analyses | |
| | | 9.5.1. | · | |
| | | 9.5.2. | Statistical consideration for Interim analyses | 83 |
| 10. | SUPP | ORTING | DOCUMENTATION AND OPERATIONAL | |
| | CONS | IDERATI | ONS | 83 |
| | 10.1. | | x 1: Regulatory, ethical, and study oversight considerations | |
| | | 10.1.1. | Regulatory and ethical considerations | |
| | | 10.1.2. | Financial disclosure | 84 |
| | | 10.1.3. | Informed consent process | 84 |
| | | 10.1.4. | Data protection | 85 |
| | | 10.1.5. | Committees structure | 85 |
| | | 10.1.6. | Dissemination of clinical study data | 86 |
| | | 10.1.7. | Data quality assurance | |
| | | 10.1.8. | Source documents | |
| | | 10.1.9. | Study and site start and closure | |
| | | | Publication policy | |
| | 10.2. | | x 2: Clinical laboratory tests | |
| | | 10.2.1. | | 89 |
| | | 10.2.2. | , | |
| | | | volunteers enrolled in preventive vaccine clinical trials | 90 |
| | 10.3. | | x 3: AEs and SAEs: Definitions and procedures for | |
| | | | g, evaluating, follow-up, and reporting | |
| | | 10.3.1. | Definition of AE | |
| | | 10.3.2. | Definition of SAE | |
| | | 10.3.3. | Solicited events | |
| | | 10.3.4. | Unsolicited AE | 95 |
| | | 10.3.5. | Recording, assessment and follow-up of AE, SAE, AESIs and pregnancies | 05 |
| | | | 10.3.5.1. AE, SAE and AESI recording | |
| | | | 10.3.5.2. Assessment of intensity | |
| | | | 10.3.5.3. Assessment of intensity | |
| | | | 10.3.5.4. Assessment of outcomes | |
| | | | 10.0.0.T. A336331116111 01 0016011163 | 50 |

# 219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| | | | 1 Totocol Amendment 5 Tina |
|---|---|---|---|
| | | • | s, SAEs, AESIs, pregnancies |
| | | or any other eve | nts of interest99 |
| | | 10.3.5.6. Updating of SAE | , AESI and pregnancy |
| | | information after | removal of write access to the |
| | | participant's eCF | RF100 |
| | | | Es, AESIs and pregnancies100 |
| | 10.4. | Appendix 4: Contraceptive guidance | |
| | | information | |
| | | 10.4.1. Definitions | 101 |
| | | | 101 |
| | | | men not considered as |
| | | | CBP (WONCBPs)101 |
| | | | 101 |
| | 10.5 | | tory103 |
| | 10.0. | Appoint A. Frotocol amonamont mo | 100 |
| 11. | REFE | RENCES | 106 |

# 219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | SoA | 28 |
| Table 2 | Intervals between study visits | 31 |
| Table 3 | Study objectives, endpoints and estimands | 34 |
| Table 4 | Part A study groups, interventions, and blinding | 37 |
| Table 5 | Part B study groups, interventions, and blinding | 37 |
| Table 6 | Part A study interventions administered | 43 |
| Table 7 | Part B study interventions administered | 44 |
| Table 8 | Contact information for emergency unblinding | 46 |
| Table 9 | Biological samples | 52 |
| Table 10 | Laboratory assays | 53 |
| Table 11 | Immunological read-outs | 54 |
| Table 12 | Study holding rules | 59 |
| Table 13 | Timeframes for collecting and reporting of safety information | 64 |
| Table 14 | List of pIMDs | 67 |
| Table 15 | Timeframes for submitting SAE, AESI, pregnancy and other events reports to CRO | 75 |
| Table 16 | Contact information for reporting SAEs, AESIs, pregnancies and study holding rules | 76 |
| Table 17 | Analysis sets | 79 |
| Table 18 | Protocol required safety laboratory assessments | 89 |
| Table 19 | Toxicity grading scales for biochemistry parameters evaluated in the current study* | 90 |
| Table 20 | Toxicity grading scales for hematology parameters evaluated in the current study* | 91 |
| Table 21 | Solicited administration site events | 94 |
| Table 22 | Solicited systemic events | 94 |
| Table 23 | Intensity scales for solicited events | 97 |

| | | 219112 (MRNA CLINRES-001) |
|---|---|---|
| | | Protocol Amendment 3 Final |
| Table 24 | Highly effective contraceptive methods | 102 |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design overview | 26 |
| Figure 2 | Probability of not meeting holding rules 1 and 2 for 8 participants per study group | 61 |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

Ab Antibody

AE Adverse event

AESI Adverse event of special interest

ANCOVA Analysis of covariance

AST Aspartate aminotransferase

BMI Body mass index

CFR Code of federal regulations

CI Confidence interval

CIOMS Council for International Organizations of Medical Sciences

CLS Clinical laboratory sciences

CoP Correlate of protection

COVID-19 Coronavirus disease 2019

CRF Case report form

CRO Contract research organization

CSL Clinical science lead

CSR Clinical study report

ECL Electro-chemiluminescence assay

ECMO Extracorporeal membrane oxygenation

eCRF electronic Case report form

EKG Electrocardiogram

EMA European Medicines Agency

EoS End-of-study

FDA Food and Drug Administration

FiO<sub>2</sub> Fraction of inspired oxygen

## 219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

FSFV First subject first visit

FSH Follicle stimulating hormone

FTIH First time in human

GCP Good clinical practice

GMC Geometric mean concentration

GMR Geometric mean ratio

GMT Geometric mean titer

GSB Global safety board

GSK GlaxoSmithKline Biologicals SA

hCG human Chorionic gonadotropin

HIPAA Health insurance portability and accountability act

HIV Human immunodeficiency virus

HRT Hormonal replacement therapy

IB Investigator's brochure

ICF Informed consent form

ICH The International Council for Harmonisation of Technical

Requirements for Pharmaceuticals for Human Use

ICMJE International Committee of Medical Journal Editors

ICS Intracellular cytokine staining

IEC Independent ethics committee

IgG Immunoglobulin G

IMP Investigational medicinal product

INR International normalized ratio

IRB Institutional review board

IRT Interactive response technology

iSRC Internal safety review committee

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

IUD Intrauterine device

IUS Intrauterine hormone-releasing system

LNP Lipid nano particles

LSLV Last subject last visit

MAAE Medically attended adverse event

MedDRA Medical dictionary for regulatory activities

mRNA-CR vaccine SARS-CoV-2 Omicron variant S glycoprotein vaccine

N Nucleocapsid

NCT National Clinical Trial

PaO<sub>2</sub> Partial pressure of oxygen

PBMC Peripheral blood mononuclear cell

PCR Polymerase chain reaction

PI Personal information

pIMD Potential immune-mediated disease

PM Pharmacy manual

PP Per Protocol

PPD Pharmaceutical Product Development

PPS Per Protocol Set

PRAC Pharmacovigilance Risk Assessment Committee

PT Preferred term

QTL Quality tolerance limit

RNASeq RNA sequencing

RT-PCR Real-time polymerase chain reaction

S Spike

SAE Serious adverse event

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

SAP Statistical analysis plan

SARS-CoV-2 Severe acute respiratory syndrome coronavirus 2

SoA Schedule of activities

SOC System organ class

SpO<sub>2</sub> Pulse oximetry

SRT Safety review team

TC Telephone call

ULN Upper limit of normal

US United States

WBC White blood cell

WOCBP Woman of childbearing potential

WONCBP Woman of non-child-bearing potential

WT SARS-CoV2 Wuhan ancestral strain or Wild type strain

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

## **Adverse Drug Reaction:**

An adverse event where a causal relationship between a medicinal product and the adverse event is at least a reasonable possibility, i.e., the relationship cannot be ruled out.

- a. In the context of a clinical trial, an ADR can be serious or non-serious. Serious ADRs may be subject to expedited reporting if they are considered unexpected (see SUSAR definition).
- b. For marketed products, ADRs are subject to expedited reporting within the country where they are authorized

## **Adverse Event (AE):**

Any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse.

# **Auxiliary Medicinal Product (AxMP):**

Medicinal products used in the context of a clinical trial but not as investigational medicinal products, such as medicinal products used for background treatment, challenge agents, rescue medication, or used to assess end-points in a clinical trial. Auxiliary medicinal products should not include concomitant medications, that is medications unrelated to the clinical trial and not relevant for the design of the clinical trial.

#### a. Authorized AxMP:

Medicinal product authorized in accordance with Regulation (EC) No 726/2004, or in any Member State concerned in accordance with Directive 2001/83/EC, irrespective of changes to the labelling of the medicinal product.

Safety reporting with regard to auxiliary medicinal products shall be made in accordance with Chapter 3 of Title IX of Directive 2001/83/EC.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

b. Unauthorized AxMP:

Medicinal product not authorized in accordance with Regulation (EC) No 726/2004.

Safety reporting for unauthorized auxiliary medicinal products will follow the same processes and procedures as SUSAR safety reporting

**Background treatment:** 

Type of medicinal product administered to each of the clinical trial participant, regardless of randomization group, to treat the indication that is the object of the study. Background treatment is generally considered to be the current standard care for the particular indication. In these trials, the IMP is given in addition to the background treatment and safety efficacy are assessed. The protocol may require that the IMP plus the background treatment is compared with an active comparator or with placebo plus background treatment.

**Blinding:** 

A procedure in which 1 or more parties to the study are kept unaware of the intervention assignment in order to reduce the risk of biased study outcomes. The level of blinding is maintained throughout the conduct of the study, and only when the data are cleaned to an acceptable level of quality will appropriate personnel be unblinded or when required in case of a serious Aes

In an observer-blind study, the participant, the site and sponsor personnel involved in the clinical evaluation of the participants are blinded while other study personnel may be aware of the treatment assignment.

**Challenge agents:** 

A product given to trial participants to produce a physiological response that is necessary before the pharmacological action of the IMP can be assessed.

Co-administered (concomitant) products:

A product given to clinical trial participants as required in the protocol as part of their standard care for a condition which is not the indication for which the IMP is being tested and is therefore not part of the objective of the study.

**Comparator:** 

Any product used as a reference (including placebo, marketed product, GSK or non-GSK) for an investigational product being tested in a clinical trial. This is any product that is being used to assess the safety, efficacy, or other measurable value against the test product (IMP).

07 Feb 2024

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

**eDiary:** Electronically registered patient data and automated data

entries on, for example, a handheld mobile device, tablet

or computer.

Eligible: Qualified for enrollment into the study based upon strict

adherence to inclusion/exclusion criteria.

**Enrollment:** The process of registering a participant into a clinical

study by assigning participant identification number

after signing the ICF.

**Essential documents:** Documents which individually and collectively permit

evaluation of the conduct of a study and the quality of

the data produced.

eTrack: GSK's tracking tool for clinical studies.

**Evaluable:** Meeting all eligibility criteria, complying with the

procedures defined in the protocol, and, therefore,

included in the per protocol analysis.

**Immunological CoP:** A correlate of risk that has been validated to predict a

certain level of protection from the targeted endpoint.

**Intervention:** Term used throughout the clinical study to denote a set

of investigational product(s) or marketed product(s) or placebo intended to be administered to a participant.

**Intervention number:** A number identifying an intervention to a participant,

according to intervention allocation.

**Investigational Product:** A pharmaceutical form of an active substance or placebo

being tested or used as a reference in a clinical trial,

including products already with a marketing

authorization but used or assembled (formulated or packaged) in a way different from the authorized form, or when used for an unauthorized indication, or when used to gain further information about the authorized

form.

**Investigational vaccine:** A pharmaceutical form of an active ingredient being

tested in a clinical study, including a product with a marketing authorization when used in a way different

from the approved form, or when used for an

unapproved indication, or when used to gain further

information about an approved use.

Synonym: IMP

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

**Investigator:** A person responsible for the conduct of the clinical

study at a study site. If a study is conducted by a team of individuals at a study site, the investigator is the

responsible leader of the team and may be called the

principal investigator.

The investigator can delegate study-related duties and functions conducted at the study site to qualified individual or party to perform those study-related duties

and functions.

Medicinal products used to assess end-points:

A product given to the participant in a Clinical Trial as a tool to assess a relevant clinical trial endpoint; it is not being tested or used as a reference in the clinical trial.

**Participant:** Term used throughout the protocol to denote an

individual who has been contacted to participate or who participates in the clinical study as a recipient of the study intervention (vaccine(s)/product(s)/control).

Synonym: subject

**Participant number:** A unique identification number assigned to each

participant who consents to participate in the study.

**Placebo:** An inactive substance or treatment that looks the same

as, and is given in the same way as, an active drug or

intervention/treatment being studied.

**Randomization:** Process of random attribution of intervention to

participants to reduce selection bias.

**Rescue medication:** Medicines identified in the protocol as those that may be

administered to the participants when the efficacy of the IMP is not satisfactory, or the effect of the IMP is too great and is likely to cause a hazard to the patient, or to

manage an emergency situation.

**Solicited event:** Events to be recorded as endpoints in the clinical study.

The presence/occurrence/intensity of these events is actively solicited from the participant or an observer during a specified follow-up period following study

intervention administration.

**Source data:** All information in original records and certified copies

of original records of clinical findings, observations, or other activities in a clinical study necessary for the reconstruction and evaluation of the study. Source data are contained in source documents (original records or

certified copies).

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

**Source documents:** 

Original legible documents, data, and records (e.g. hospital records, clinical and office charts, laboratory notes, memoranda, participants' diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate copies, microfiches, photographic negatives, microfilm or magnetic media, x-rays, participant files, and records kept at the pharmacy, laboratories and at medicotechnical departments involved in the clinical study).

**Standard of Care:** 

Medicine(s) for a specific indication, or a component of the standard care for a particular medical indication, based on national and/or international consensus; there is no regulatory significance to this term.

Products/regimens considered standard of care may differ country to country, depending on consensus in individual countries

**Study intervention:** 

Any investigational or marketed product(s) or placebo intended to be administered to a participant during the study.

**Study monitor:** 

An individual assigned by the sponsor and responsible for assuring proper conduct of clinical studies at 1 or more investigational sites.

**SUSAR:** 

Suspected Unexpected Serious Adverse Reaction; in a clinical trial, a serious adverse reaction that is considered unexpected, i.e., the nature or severity of which is not consistent with the reference safety information (e.g., Investigator's Brochure for an unapproved investigational medicinal product). All adverse drug reactions (ADRs) that are both serious and unexpected are subject to expedited reporting.

**Telemedicine:** 

The use of electronic information and telecommunications technologies (both video-based and audio-only) to facilitate remote health care delivery, patient and professional health-related education, public health and health administration.

**Unsolicited AE:** 

Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited AE.

# 1. PROTOCOL SUMMARY

# 1.1. Synopsis

**Rationale:** GSK is developing a novel mRNA vaccine platform where the SARS-CoV-2 Omicron variant S glycoprotein will be used as an antigen model (hereafter referred to as mRNA-CR vaccines). This mRNA vaccine platform development includes several mRNA constructs (mRNA-CR-XX) currently under development that will be progressing into clinical research in humans.

**Objectives, endpoints and estimands:** This exploratory, FTIH study is to evaluate the safety, reactogenicity and immune responses of the mRNA-CR-04 vaccine construct when administered in healthy adults previously vaccinated with SARS-CoV-2 mRNA vaccines. For details on objectives, endpoints and estimands, refer to Section 3.

Overall design: This will be a Phase 1, observer-blind, randomized, placebo-controlled, multicenter, dose-escalation study evaluating in Part A of the study, 3 doses ( $10 \mu g$ ,  $30 \mu g$ , and  $100 \mu g$ ) of the mRNA-CR-04 (Omicron BA.5 strain) vaccine. Approximately 72 participants will be enrolled with 24 participants per group (Group 1, Group 2 and Group 3). Within each group, participants will be randomly assigned in a 3:1 ratio to receive:

- investigational mRNA-CR-04 vaccine (SPK001-AC01 mRNA-LNP) or
- saline placebo.

For each group, 8 sentinel participants will first be enrolled and vaccinated. Enrollment of participants in Group 1 and Group 2 will be done in parallel with the first participant to be enrolled in Group 1. Only if no safety signal is observed, vaccination of the non-sentinel participants in that group will continue. If no safety signals observed in sentinel participant in Group 1 and Group 2, enrollment, and vaccination of the sentinel participants in Group 3 will be initiated. Refer to Section 4.1 and Figure 1 for more details on the study design.

Part B of the study will commence only after all Part A participants have completed their Day 15 study visits and the Day 15 interim analysis is completed. In Part B, 2 doses (3  $\mu$ g and 10  $\mu$ g) of the mRNA-CR-04 (Omicron BA.5 strain) vaccine will be evaluated. Approximately 42 participants will be enrolled in parallel in Part B and there will be no sentinel participants. Part B participants will be randomly assigned in a 3:3:1 ratio to receive:

- 3 µg investigational mRNA-CR-04 vaccine (SPK001-AC01 mRNA-LNP) or
- 10 µg investigational mRNA-CR-04 vaccine (SPK001-AC01 mRNA-LNP) or
- saline placebo.

**Data Monitoring/Other committees:** Safety monitoring and safety data review will be performed by a GSK SRT (blinded data review until Part A Day 15 interim analysis, unblinded data review subsequently) and a GSK iSRC (unblinded data review). Safety holding rules and safety monitoring are presented in Section 8.3.7.

# 1.2. Schema

This is an exploratory, FTIH, observer-blind, randomized, multicenter, controlled study.

In Part A of the study, three doses ( $10 \mu g$ ,  $30 \mu g$ , and  $100 \mu g$ ) of the mRNA-CR-04 vaccine will be evaluated. Approximately 72 eligible healthy adults, 18 to 49 years, inclusive, will be enrolled with 24 participants per group (Group 1, Group 2 and Group 3). Within each group, participants will be randomly assigned in a 3:1 ratio:

- 18 participants will receive the investigational mRNA-CR-04 vaccine and
- 6 participants will receive a saline placebo (sodium chloride [NaCl] isotonic solution [0.9%]).

In Part B of the study, two doses (3  $\mu$ g and 10  $\mu$ g) of the mRNA-CR-04 vaccine will be evaluated. Approximately 42 eligible healthy adults, 18 to 49 years, inclusive, will be enrolled in Part B and will be randomly assigned in a 3:3:1 ratio:

- 18 participants will receive 3 μg of the investigational mRNA-CR-04 vaccine and
- 18 participants will receive 10 μg of the investigational mRNA-CR-04 vaccine and
- 6 participants will receive a saline placebo (sodium chloride [NaCl] isotonic solution [0.9%]).

Study duration for all the participants will be approximately 6 months, and they will be evaluated for safety, reactogenicity and immunogenicity. Safety monitoring and safety data review will be performed by a GSK SRT (blinded data review until Part A Day 15 interim analysis, unblinded data review subsequently) and a GSK iSRC (unblinded data review).

Overview of study design is presented in Section 4.1. Safety holding rules and safety monitoring are presented in Section 8.3.7.

Figure 1 Study design overview



219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

CMI: Cell-mediated immunity; D: Day; M: Month; mRNA: mRNA-CR-04 vaccine; n: Number of participants; SE: Solicited events; TC: Telephone call; V: Visit.

\* TC1 D2 only for sentinel participants in each group. \*\* The first participant is to be enrolled in Group 1. In addition to the defined intervals between doses within each group, an interval of at least 60 minutes will be maintained between the vaccination of sentinel participants across Group 1 and Group 2. \*\*\* TC1 review will be performed by the SRT on blinded data.

# 1.3. Schedule of Activities (SoA)

# Table 1 SoA

| Type of contact | Screening | Visit 1 | TC1* | Visit 2 | Visit 3 | Visit 4 | TC2 | Visit 5 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time points | period | D1 | D2 | D8 | D15 | D31 | М3 | M6 | Fault II | llaaabadulad | Unscheduled | |
| Window (D) | D-14 to -1 | 0 | 0 | +2 | ±2 | ±3 | ±5 | ±7 | Early termination | Unscheduled COVID-19+ | cardiac | Notes |
| Assessment and sampling time | Pre-Vacc | Pre- | Post- | Post- | Post- | Post- | Post- | Post- | termination | COAID-18. | evaluation | |
| points | | Vacc | Vacc | Vacc | Vacc | Vacc | Vacc | Vacc | | | | |
| Screening | | | | | | | | | | | | |
| Informed consent | • | | | | | | | | | | | Section 10.1.3 |
| Inclusion/exclusion criteria | • | | | | | | | | | | | Section 5.1 and |
| | • | | | | | | | | | | | Section 5.2 |
| Demography | • | | | | | | | | | | | Section 8.1.1 |
| Medical history | • | | | | | | | | | • | | Section 8.1.2 |
| Vaccination history | • | | | | | | | | | | | Section 8.1.2 |
| Physical examination | • | •*** | | | | | | | | • | | Section 8.3.1 |
| Vital signs measurement | • | •*** | | | | | | | | • | | Section 8.3.1 |
| Body temperature | | | | | | | | | | | | Section 8.3.2 |
| | | | | | | | | | | | | The preferred |
| | | | | | | | | | | | | location for |
| | | | | | | | | | | | | measuring |
| | • | •*** | | | | | | | | • | | temperature will be: |
| | | | | | | | | | | | | oral. |
| | | | | | | | | | | | | Fever is defined as |
| | | | | | | | | | | | | body temperature |
| | | | | | | | | | | | | ≥38°C/100.4°F. |
| Pregnancy test ** | • | • | | | | | | | | | | Section 8.3.3 |
| Study intervention | | | | | | | | | | | | |
| Participant randomization | | • | | | | | | | | | | Section 6.3 |
| Vaccine administration | | • | | | | | | | | | | Section 6.1 |
| Initiation of eDiary | | • | | | | | | | | | | Section 8.1.3 |

219112 (MRNA CLINRES-001)
Protocol Amendment 3 Final

| Type of contact | Screening | Visit 1 | TC1* | Visit 2 | Visit 3 | Visit 4 | TC2 | Visit 5 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time points | period | D1 | D2 | D8 | D15 | D31 | М3 | M6 | Fambr | Hannaha dula d | Unscheduled | |
| Window (D) | D-14 to -1 | 0 | 0 | +2 | ±2 | ±3 | ±5 | ±7 | Early Unscheduled termination COVID-19+ | cardiac | Notes | |
| Assessment and sampling time | Pre-Vacc | Pre- | Post- | Post- | Post- | Post- | Post- | Post- | termination | COAID-18. | evaluation | |
| points | | Vacc | Vacc | Vacc | Vacc | Vacc | Vacc | Vacc | | | | |
| Laboratory assessment | | | | | | | | | | | | |
| SARS-CoV-2 N protein serology | | • | | | • | • | | • | • | | | Section 8.2.1 |
| SARS-CoV-2 RT-PCR | • | • | | • | • | | | | | • | | Section 8.2.1 |
| nasopharyngeal swab) | | | | | | | | | | | | 0 |
| Blood sample for binding IgG | | • | | | • | • | | • | • | | | Section 8.2.1 |
| Blood sample for neutralization | | • | | | • | • | | • | • | | | Section 8.2.1 |
| Blood sample for PBMC ICS assay<br>preparation | | • | | | • | • | | • | • | | | Section 8.2.1 |
| Safety assessments | | | | | | <b>B</b> . | | u. | | | | |
| Hematology and serum chemistry | • | • | | • | • | | | | | | • | Section 8.3.6 |
| Cardiac troponin I | • | | | • | | | | | | | • | Section 8.2.1 |
| Record any concomitant medication/vaccination | • | • | | • | • | • | • | • | • | • | | Section 6.8 |
| Record solicited AEs in eDiary (up o 7 days after vaccination) | | 0 | | 0 | | | | | | | | Section 8.4 |
| Record unsolicited AEs (up to 30 days after vaccination) | | • | • | • | • | • | | | | | | Section 8.4 |
| Reporting of SAEs, MAAEs, AESI including COVID-19), and pregnancies | | • | • | • | • | • | • | • | • | • | • | Section 8.4 |
| Recording of SAEs related to | | | | | | | | | | | | Section 8.4 |
| tudy participation, or to a<br>oncurrent GSK<br>nedication/vaccine | • | • | • | • | • | • | • | • | • | • | • | |
| EKG | • | | | • | | | | | | | • | Section 8.3.4 |
| - | • | | | • | | | | <del> </del> | | | • | 3600011 0.3.4 |
| Study Conclusion | | | | | | | | • | • | | | |

AE: Adverse event; AESI: Adverse events of special interest; D: Day; eCRF: electronic Case report form; eDiary: electronic Diary card; EKG: Electrocardiogram; GSK: GlaxoSmithKline Biologicals SA; ICS: Intracellular cytokine staining; IgG: Immunoglobulin G; M: Month; MAAE: Medically attended adverse event; N: Nucleocapsid; PBMC: Peripheral blood mononuclear cell; pIMD: potential Immune-mediated disease; RT-PCR: Real-time polymerase chain reaction; SAE: Serious adverse event; TC: Telephone call; Vacc: Vaccination.

219112 (MRNA CLINRES-001)
Protocol Amendment 3 Final

Diagnosis of COVID-19 should be made in accordance with the World Health Organization [WHO, 2023] case definitions. Cases should be reported as AESIs or SAEs, and routine procedures for recording, evaluation, follow-up, and reporting of AESIs, and SAEs should be followed in accordance with the protocol-defined time periods.

- \* TC1 is only for sentinel participants in each group in Part A.
- \*\* Female participants of childbearing potential must perform a urine pregnancy test before the administration of the study intervention. For screening, if time allows, a serum pregnancy test can be done, in place of the urine pregnancy test, as per local requirements.
- \*\*\* Physical examination, vital signs, and body temperature measurement at D1 will occur before vaccination.
- + Procedures apply to both suspected and convalescent visits for COVID-19.

Note: The double-line border following D15 indicates the analyses which will be performed on all data (i.e., data that are as clean as possible) obtained up to D15.

- Is used to indicate a study procedure that requires documentation in the individual eCRF.
- o Is used to indicate a study procedure that requires documentation in the eDiary.

Table 2 Intervals between study visits

| Interval | Planned visit interval | Allowed interval range |
|---|---|---|
| Screening → Visit 1 (D1) | 1-14 days* | 1-14 days |
| Visit 1 (D1) → TC1 (D2) | 1 day | 1 day |
| Visit 1 (D1) → Visit 2 (D8) | 7 days | 7-9 days |
| Visit 1 (D1) → Visit 3 (D15) | 14 days | 12-16 days |
| Visit 1 (D1) → Visit 4 (D31) | 30 days | 27-33 days |
| Visit 1 (D1) → TC2 (M3) | 90 days | 85-95 days |
| Visit 1 (D1) → Visit 5 (M6) | 180 days | 173-187 days |

D: Day; M: Month; PCR: Polymerase chain reaction; TC: Telephone call.

#### 2. INTRODUCTION

# 2.1. Study rationale

As part of developing a novel mRNA vaccine platform, GSK selected the SARS-CoV-2 S glycoprotein as a model antigen (mRNA-CR vaccine). This is an exploratory, FTIH, observer-blind, randomized, controlled study, evaluating various doses of mRNA-CR-04 in individuals who have previously received:

• 2-dose primary series and booster dose(s) of an authorized or licensed mRNA COVID-19 vaccine (only Moderna or Pfizer vaccines) with the last booster dose administered at least 6 months or more prior to screening.

The safety, reactogenicity and immunogenicity of the mRNA-CR-04 vaccine administered in healthy adults previously vaccinated with a SARS-CoV-2 mRNA vaccine will be evaluated. The decision to move this mRNA construct and dose forward for the development of vaccines for a specific disease will be based on safety, reactogenicity, and immunogenicity profiles of the construct compared to the current standard of care.

# 2.2. Background

Due to the ongoing impact of COVID-19, there is a need for vaccines to provide protection against COVID-19 caused by SARS-CoV-2 variants of concern. As of 03 March 2023, more than 675 million cases have been reported worldwide, leading to more than 6.8 million deaths [Mathieu, 2023]. To date, there are multiple licensed or conditionally approved vaccines available that rely on a variety of vaccine technologies.

With the surge in Omicron predominance worldwide, its greater transmissibility, and a higher risk of SARS-CoV-2 reinfection with Omicron [Garcia-Beltran, 2021; Zhou, 2021], it is reasonable to anticipate an urgent need for booster vaccines to expand immunity against Omicron and additional future variants of concern. Bivalent boosters encoding Omicron BA.4/5 and the ancestral S protein sequences, followed by monovalent boosters encoding XBB.1.5 since 11 September 2023, have been authorized

<sup>\*</sup> Visit 1 should take place no longer than 14 days after the Screening visit. All screening procedures, except the SARS-CoV-2 PCR test, need to be performed within 14 days of Visit 1 (see Section 8.1 and Section 8.3). A SARS-CoV-2 PCR test needs to be performed within 7 days of Visit 1. When applicable, a sample may be collected for repeat testing at any time (but only once to assess eligibility) before Visit 1. Only laboratory results from the repeat test, if it occurs, will be taken into consideration. The participant can only be assigned to a study intervention group once the investigator receives the results and confirms eligibility.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

for all doses administered to individuals 6 months of age and older [FDA, 2023a; FDA, 2023b].

Please refer to the current IB for information regarding preclinical studies of mRNA-CR-04 vaccine.

## 2.3. Benefit/risk assessment

Detailed information about the known and expected benefits and risks and expected AEs of mRNA-CR-04 vaccine can be found in the IB.

With any vaccine, administration site (e.g., pain, swelling, redness) and systemic (e.g., fever, fatigue, headache, myalgia) post-dosing events may occur within the first 3 days of study intervention administration, and are anticipated to be resolved within a few days of onset.

Syncope can occur following an injectable vaccine or even before any vaccination as a vasovagal response to the needle injection. Similarly, hypersensitivity reactions may also occur.

Currently, there are no identified preclinical risks for the investigational mRNA-CR-04 vaccine. However, the following important potential risks and mitigation strategies have been defined for this vaccine:

#### Risk Assessment

| Important/potential/risk of clinical significance | Summary of data/rationale for risk | Mitigation strategy |
|---|---|---|
| All study vaccines | | |
| Hypersensitivity reactions including allergic reactions such as anaphylaxis | Acute allergic reactions such as a rare case of anaphylactic event may occur with any vaccine - administration. These are serious, but rare occurrences estimated in the range of 1 to 10 cases per million of vaccinations, depending on the vaccine studied [Rüggeberg, 2007]. | A history of hypersensitivity or severe allergic reaction (including anaphylaxis) is an exclusion criterion for study participation and a contraindication to vaccination. The onset of vaccine-related allergic symptoms is typically quite prompt. To treat participants with a serious allergic vaccination reaction, all participants will need to remain under observation (i.e., visibly followed; no specific procedure) at the study site for at least 60 minutes after vaccination. Participants will be instructed to contact the study site immediately for occurrence of any possible hypersensitivity reaction within 1 day following study intervention administration. |
| Bleeding following intramuscular injection | As with other intramuscular injections, study intervention should be given with caution in individuals with bleeding disorders, such as hemophilia or on anticoagulant | To minimize the risk of bleeding, study intervention should be given with caution in individuals with thrombocytopenia or any coagulation disorder. |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Important/potential/risk of clinical significance | Summary of data/rationale for risk | Mitigation strategy |
|---|---|---|
| | therapy, to avoid the risk of hematoma following the injection. | Participants with any medical condition that in judgment of the investigator would make intramuscular injection unsafe will be excluded from study enrollment. |
| mRNA-CR-04 vaccine | | |
| Myocarditis/pericarditis | Myocarditis/pericarditis are considered as an important identified risk for marketed mRNA COVID-19 vaccines [EMA, 2021a; EMA, 2021b; FDA, 2021a; FDA, 2021b] The estimated reporting rates of myocarditis in younger adults [25- to 29-year old] following the first and the second doses of BNT162b2 vaccine were 0.7 and 5.7 per 100 000, respectively and following the first and the second doses of mRNA-1273 vaccine were 1.8 and 11.2 per 100 000, respectively [CDC, 2021]. The same reporting trend was observed following booster mRNA vaccination, except for age, with most cases reported in older adults [ACIP, 2021]. | Participants at increased risk of myocarditis/pericarditis or with medical history of myocarditis/pericarditis are excluded from study enrollment. Participants will also be instructed (via informed consent form) to be alert for symptoms of myocarditis/pericarditis and immediately contact the site if any of these symptoms occur. Participants will be tested for cardiac troponin I and undergo EKG at the screening and on D8 after study intervention administration. Participants will receive close medical supervision and medical assessments (e.g., laboratory testing) during the study. Moreover, myocarditis/pericarditis will be collected as an AESI and adjudicated (refer to Section 8.3.8, Section 8.4.4 and Section 10.3.5) |
| Vaccine-associated disease enhancement | Enhanced disease following vaccination has been observed in pre-clinical or clinical studies with various vaccines (e.g., RSV, Dengue, SARS) and the mechanism is poorly understood [Peeples, 2020]. While there are literature reports of enhanced disease in animals vaccinated with previous SARS vaccines, some other reports fail to see this effect. | During informed consent process, participants will be informed of this theoretical risk and asked to report any symptoms consistent with COVID-19 and/or for which they received medical attention at any point during the study. Any suspected, probable, or confirmed case of COVID-19 (regardless of severity) is an AESI; and will be captured and described (refer to Section 8.4.4 and Section 10.3.5) |

AESI: Adverse event of special interest; EKG: Electrocardiogram; D: Day; RSV: Respiratory syncytial virus; SARS: Severe acute respiratory syndrome.

#### **Benefit assessment**

Participants may gain information about their general health status through medical evaluations/assessments associated with this study (i.e., physical examinations and blood testing [hematology and biochemistry data]).

## **Overall Benefit: Risk conclusion**

The investigational mRNA-CR-04 vaccine is currently in an early stage of clinical development and vaccine efficacy, immunogenicity, and safety have not yet been demonstrated in humans.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Based on the available data for currently authorized/licensed mRNA COVID-19 vaccines, some potential risks have been defined. Appropriate safety monitoring and evaluation methodologies are in place to quickly identify any such events, should they occur.

Thus, while the benefit of this vaccine has not yet been proven, the anticipated potential risks for the mRNA-CR-04 vaccine are justified by the anticipated potential benefits.

# 3. OBJECTIVES, ENDPOINTS, AND ESTIMANDS

Table 3 Study objectives, endpoints and estimands

| | Objective(s) | Endpoints/Estimands |
|---|---|---|
| | Primary | |
| • | To evaluate the safety and reactogenicity of investigational mRNA-CR-04 vaccine up to D31 | <ul> <li>Solicited administration site events and systemic events during the 7-day follow-up period after study vaccine administration (day of study vaccine administration and 6 subsequent days);</li> <li>Unsolicited AEs during the 30-day follow-up period after study vaccine administration (day of study vaccine administration and 29 subsequent days);</li> </ul> |
| | | <ul> <li>Any hematological and biochemical laboratory abnormality during the 15-day follow-up period after study vaccine administration (day of study vaccine administration and 14 subsequent days);</li> <li>MAAEs; SAEs; AESIs* up to D31.</li> </ul> |
| | Seconda | ry Safety |
| • | To assess safety of investigational mRNA-CR-04 vaccine from study vaccine administration up to study conclusion. | MAAEs; SAEs; AESIs* up to study conclusion (M6). |
| | Secondary Immunogenicity | |
| • | To evaluate the Ab functionality (neutralizing capacity induced by the mRNA-CR-04 vaccine against vaccine encoded SARS-CoV-2 and WT strains) up to study conclusion. | <ul> <li>Neutralizing titer GMTs against pseudovirus bearing S protein from vaccine encoded SARS-CoV-2 and WT strains at each collection timepoint (D1, D15, D31, M6).</li> <li>GMR from baseline (D1) of neutralizing titer against pseudovirus bearing S protein from vaccine encoded SARS-CoV-2 and WT strains at each collection timepoint.</li> <li>Vaccine response rate based on neutralizing titers against vaccine encoded SARS-CoV-2 and WT strains at each collection timepoint.</li> </ul> |
| | Terti | ary |
| • | To describe serum-binding antibody (IgG) responses induced by the mRNA-CR-04 vaccine specific for vaccine encoded SARS-CoV-2 and WT strains S protein up to study conclusion. | GMCs of binding IgG Ab specific for S protein encoded by the vaccine SARS-CoV-2 and WT strains at each timepoint (D1, D15, D31, M6). GMR from baseline of binding IgG Ab specific for S protein encoded by the vaccine SARS-CoV-2 and WT strains S proteins at each timepoint. Seroresponse rates based on binding IgG concentrations specific for S protein encoded by the vaccine SARS-CoV-2 and WT strains S protein at each timepoint. |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Objective(a) | Endnoints/Estimonds |
|---|---|
| Objective(s) | Endpoints/Estimands |
| To describe cell-mediated immune responses induced by the mRNA-CR-04 vaccine up to study conclusion. | <ul> <li>Frequency of CD4+/CD8+ T-cells specific for S protein encoded by the vaccine SARS-CoV-2 and WT strains measured by intracellular cytokine staining assay at each time point (D1, D15, D31, M6).</li> <li>Cellular immune responses including, but not limited to Th1 and Th2 profiles as determined by flow cytometry using ICS at each time point (D1, D15, D31, M6).</li> </ul> |
| To describe the incidence of confirmed symptomatic and asymptomatic SARS-CoV-2 infection. | <ul> <li>Percentage of laboratory-confirmed (N protein seroconversion) asymptomatic SARS-CoV-2 infection at each time point (D1, D15, D31, M6).</li> <li>Percentage of laboratory-confirmed (RT-PCR) symptomatic SARS-CoV-2 infection at screening, D1, D8, D15, as well as at unscheduled visits.</li> </ul> |
| To evaluate the genetic sequence of SARS-CoV-2 variant S protein in confirmed (RT-PCR) SARS-CoV-2 positive participants. | <ul> <li>Comparison of SARS-CoV-2 S protein genetic sequence of viral isolates (when available) to the vaccine mRNA sequence</li> <li>Identification of SARS-CoV-2 variants.</li> </ul> |
| To further characterize the humoral response<br>(including, but not limited to functionality of<br>antibodies) and cellular response, specific for the<br>vaccine encoded SARS-CoV-2, WT and other<br>relevant strains. | <ul> <li>S-specific responses at D1, D15, D31, M6</li> <li>Other read-outs may be performed if deemed necessary.</li> </ul> |

Ab: Antibody; AE: Adverse event; AESI: Adverse events of special interest; D: Day; GMR: Geometric mean ratio; GMT: Geometric mean titer; ICS: intracellular cytokine staining; IgG: Immunoglobulin G; M: Month; MAAE: Medically attended adverse events; N: Nucleocapsid; pIMD: potential Immune-mediated disease; RT-PCR: Real-time polymerase chain reaction; S: Spike; SAE: Serious adverse event; VAED: Vaccine associated enhanced disease; WT: Wild type.

\*AESI include pIMDs, myocarditis/pericarditis, virologically confirmed COVID-19 cases and anaphylaxis or severe hypersensitivity within 24 hours after study vaccination (Section 8.4.4).

Details related to attributes of estimands covering intercurrent events and strategies, population, treatment condition, and population level summary will be provided in SAP.

#### 4. STUDY DESIGN

# 4.1. Overall design

**Experimental Design:** Phase 1, observer-blind, randomized, placebo-controlled, multicenter, dose-escalation study to evaluate in Part A of the study, 3 doses ( $10~\mu g$ ,  $30~\mu g$ , and  $100~\mu g$ ) of the mRNA-CR-04 (Omicron BA.5 strain) vaccine (Figure 1) in 3 groups (Group 1, Group 2 and Group 3) (Table 4). Part B of the study will commence only after all Part A participants have completed their Day 15 study visits and the Day 15 interim analysis is completed. In Part B (Table 5), 2 doses ( $3~\mu g$  and  $10~\mu g$ ) of the mRNA-CR-04 (Omicron BA.5 strain) vaccine will be evaluated (Figure 1). The study will be conducted in the United States (US).

**Duration of the study:** Approximately 6 months after dosing.

**Sentinel dosing**: In Part A of the study, each group will have 8 sentinel participants (6 receiving the mRNA-CR-04 vaccine and 2 receiving a placebo) who will be enrolled and

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

vaccinated in each group. The first and second sentinel participant in each group will be vaccinated and followed-up for 24 hours before the next sentinel participant can be vaccinated. Vaccination of the remaining sentinel participants in the same group will then continue with an interval of at least 60 minutes between participants. Additionally, an interval of at least 60 minutes will be maintained between the vaccination of sentinel participants across groups.

**Dose-escalation:** In Part A of the study, enrollment of participants in Group 1 and Group 2 will be done in parallel with the first participant to be enrolled in Group 1. All safety data up to Day 8 post-vaccination from sentinel participants in both groups will be reviewed by the iSRC (unblinded review). The iSRC members will determine whether any of the pre-defined holding rules are met or if there is any other safety signal. If no safety signal is observed, vaccination of the non-sentinel participants in that group will continue. If no safety signal observed from sentinel participants in Group 1 and Group 2, enrollment and vaccination of the sentinel participants in Group 3 will be initiated. In Part B, irrespective of dose, all participants in the three study groups will be enrolled in parallel.

**Safety Data:** Safety data will be collected for 6 months post-vaccination. Solicited AEs will be collected for 7 days (day of vaccination and 6 subsequent days) and unsolicited AEs will be collected up to Day 31. MAAEs, SAEs, pIMDs, and AESIs will be collected for the duration of the study. In addition to the review of unblinded data by iSRC, blinded data until Part A Day 15 interim analysis, and unblinded data subsequently, will be regularly reviewed by the SRT. For more detailed information, refer to Section 8.3 and Section 8.4.

For the vendors that will perform key study-related duties or activities, please refer to the separate list of vendors.
Table 4 and Table 5 describe the Part A and Part B study groups, interventions, and blinding, respectively.

Table 4 Part A study groups, interventions, and blinding

| Study | Number of | Age (Min- | Study intervention(s) | /vaccine(s) mode of | Blinding |
|---|---|---|---|---|---|
| groups | participants | Max years of age) | adminis | Screening→Visit 5 | |
| | 18 | 18 – 49 | mRNA-CR-04 vaccine 10 µg | Intramuscular injection into the | |
| Group 1 | Group 1 Saline placebo | | deltoid muscle,<br>preferably of the non-<br>dominant arm. | Observer-blind | |
| | 18 | 18 – 49 | mRNA-CR-04 vaccine 30 µg | Intramuscular injection into the | |
| Group 2 | 6 | 18 – 49 | Saline placebo<br>(NaCl [0.9%]) | deltoid muscle,<br>preferably of the non-<br>dominant arm. | Observer-blind |
| | 18 | 18 – 49 | mRNA-CR-04 vaccine<br>100 μg | Intramuscular injection into the | |
| Group 3 | 6 | 18 – 49 | Saline placebo<br>(NaCl [0.9%]) | deltoid muscle,<br>preferably of the non-<br>dominant arm. | Observer-blind |

NaCl: Sodium chloride.

Table 5 Part B study groups, interventions, and blinding

| Study<br>groups | Number of participants | Age (Min-<br>Max years<br>of age) | Study intervention(s) adminis | Blinding | |
|---|---|---|---|---|---|
| Part B<br>3 µg | 18 | 18 – 49 | mRNA-CR-04<br>vaccine 3 μg | Intramuscular injection into the deltoid muscle, preferably of the non-dominant arm. | Observer-blind (except sponsor) |
| Part B<br>10 µg | 18 | 18 – 49 | mRNA-CR-04<br>vaccine 10 μg | Intramuscular injection into the deltoid muscle, preferably of the non-dominant arm. | Observer-blind (except sponsor) |
| Part B<br>Placebo | 6 | 18 – 49 | Saline placebo<br>(NaCl [0.9%]) | Intramuscular injection into the deltoid muscle, preferably of the non-dominant arm. | Observer-blind (except sponsor) |

NaCl: Sodium chloride.

# 4.2. Scientific rationale for study design

To ensure maximum safety of the participants, as this will be the first time that the mRNA-CR-04 vaccine will be administered in humans, the study will follow an observer-blind design with staggered enrollment and dosing for Part A of the study, with study holding rules and close safety monitoring throughout the study as specified in Section 4.1 and Section 8.3.7. Part B of the study adds an even lower dose (3 µg) of

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

mRNA-CR-04 vaccine group to allow exploration of a wider range of vaccine doses, as well as a repeat of the Part A low dose (10  $\mu$ g) of mRNA-CR-04 vaccine group, which may assist in standardizing the new 3  $\mu$ g dose group in Part B to the earlier Part A study groups.

#### 4.3. Justification for dose

The proposed doses will be 3 μg, 10 μg, 30 μg, and 100 μg. The monovalent SARS-CoV-2 mRNA vaccines (Pfizer-BioNTech Comirnaty mRNA vaccine [FDA, 2023a] and Spikevax Moderna COVID-19 Vaccine [FDA, 2023b]) have been licensed in the US as a 2 or 3-dose primary series. Bivalent formulations of the Moderna and Pfizer-BioNTech COVID-19 vaccines encoding S protein sequences from Omicron BA.4/5 and the ancestral strain followed by monovalent boosters encoding XBB.1.5 since 11 September 2023, have been authorized for primary and booster vaccinations [FDA, 2023a; FDA, 2023b].

The maximum planned dose is  $100 \mu g$ . The rationale for evaluating doses from 3  $\mu g$  to  $100 \mu g$  is based on the following considerations:

- The optimal dose required to confer cross-protective immunity against non-Omicron variants, including new/emerging variants needs to be determined.
- Moderna has evaluated doses up to 250 μg (2-dose regimen) in their Phase 1 studies [Jackson, 2020].
- The doses of the authorized bivalent booster vaccines from Pfizer-BioNTech and Moderna are 30 μg and 50 μg, respectively. The initial starting dose of 10 μg of the mRNA-CR-04 vaccine in Part A of the study is well below these doses.

# 4.4. End-of-study definition

A participant is considered to have completed the study if he/she returns for the last visit as described in the protocol.

EoS: LSLV (Visit 5, Month 6) or date of the last testing released of the human biological samples, related to primary and secondary endpoints, whichever occurs later. EoS must be achieved no later than 8 months after LSLV. EoS cannot be before LSLV.

#### 5. STUDY POPULATION

Adherence to the inclusion and exclusion criteria specified in the protocol is essential. Deviations from these criteria are not allowed because they can jeopardize the scientific integrity, regulatory acceptability of the study or safety of the participant.

#### 5.1. Inclusion criteria

All participants must satisfy ALL the following criteria prior to dose administration:

- 1. Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.
- 2. Participants, who in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary and study procedures).
- 3. Has received 2 doses of primary series and booster dose(s) of an authorized or licensed mRNA COVID-19 vaccine (only Moderna or Pfizer vaccines) with the last booster dose administered at least 6 months or more prior to screening and has provided documentation of receiving the vaccination series (e.g., vaccination card).
- 4. Negative for SARS-CoV-2 infection by RT-PCR test at screening within 7 days prior to study vaccination.
- 5. Is a male or nonpregnant female of 18 to 49 years, inclusive, at screening.
- 6. If the participant is a WOCBP, the participant agrees to practice true abstinence or use at least 1 highly effective form of contraception for at least 30 days prior to study vaccination up to 1 month after study vaccination.
- 7. Agrees to refrain from blood or plasma donation from screening and up to 6 months after vaccination.
- 8. Is healthy or medically stable as determined by investigator judgment based on medical history, clinical laboratory tests, vital sign measurements, and physical examination findings.

#### 5.2. Exclusion criteria

The following criteria should be checked at the time of screening and on D1 prior to dose administration. The potential participant MUST NOT be included in the study if ANY exclusion criterion applies:

#### 5.2.1. Medical conditions

- 1. Has a new onset, clinically significant, abnormal biochemistry or hematology finding (defined as ≥Grade 1) at screening (participants with Grade 1 laboratory abnormalities that have been stable for at least 6 months before enrollment may be included in the study).
- 2. Has any medical disease or condition that, in the opinion of the investigator, precludes study participation. This includes any acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of the trial.
- 3. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- 4. History of myocarditis, pericarditis, second and third degree heart block or idiopathic cardiomyopathy, or presence of any medical condition that increases risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis eosinophilic granulomatosis with polyangiitis, persistent myocardial viral infection (e.g., due to enterovirus or adenovirus).
- 5. Has an acute febrile illness with a temperature ≥38.0°C or ≥100.4°F observed by the participant or at the study site within 72 hours prior to study vaccination. Participants with suspected COVID-19 symptoms (Section 8.4.4.2.2) should be excluded and referred for medical care.
- 6. Has a history of hypersensitivity or severe allergic reaction, including anaphylaxis, generalized urticaria, angioedema, and other significant reactions to any previous vaccine, or any component of the study vaccine.
- 7. Has a body mass index  $>40 \text{ kg/m}^2$ .
- 8. Has had known close contact with anyone who had a confirmed SARS-CoV-2 infection within 14 days before study vaccination.
- 9. Has a history of documented SARS-CoV-2 infection or COVID-19 within 6 months before the date of screening visit.
- 10. Has any self-reported or medically documented clinically significant medical or psychiatric condition. Significant medical conditions include, but are not limited to, the following:
  - a. Moderate or severe respiratory disease (e.g., chronic obstructive pulmonary disease, asthma).
  - b. Uncontrolled hypertension, defined as an average systolic blood pressure ≥140 mmHg or an average diastolic blood pressure ≥90 mmHg, based on an average of up to 3 blood pressure measurements.
  - c. Clinically significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease).
  - d. Neurological or neurodevelopmental conditions (e.g., Down syndrome, dementia, chronic migraine not controlled by medication, epilepsy, stroke or seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, or transverse myelitis).
  - e. Ongoing malignancy or recent diagnosis of malignancy in the last 5 years (excluding basal cell and squamous cell carcinoma of the skin).
  - f. Tuberculosis or non-tuberculosis mycobacterial infection.
  - g. Autoimmune disease, including hypothyroidism without a defined nonautoimmune cause.
  - h. Immunodeficiency of any cause, including from solid organ transplant, blood, or bone marrow transplant, or use of other immune-weakening medicine.
  - i. Type 1 or 2 diabetes mellitus regardless of disease control.
- 11. Has any of the following self-reported or medically documented risk factors for severe COVID-19:

- a. Chronic kidney disease
- b. Cerebrovascular disease
- c. Cystic fibrosis
- d. Chronic liver disease
- e. Pulmonary fibrosis

## 5.2.2. Prior/concomitant therapy

- 12. Has participated or plans to participate in another investigational study involving any investigational drug or device within 60 days or 5 half-lives, whichever is longer, before study vaccination and throughout the study.
- 13. Has received a licensed or authorized non-mRNA COVID-19 vaccine (primary series or booster dose).
- 14. Has received or plans to receive any licensed vaccine within 4 weeks before or after study vaccination. Inactivated vaccines for influenza are permitted during the study if they are administered at least 14 days before or after study vaccination.
- 15. Is planning to receive an authorized or licensed COVID-19 booster vaccination for the duration of the study (for participants who are not covered by local recommendations to receive booster per current standard of care) OR is planning to receive an authorized or licensed COVID-19 booster vaccination on or before Day 31 of the study (for participants covered by local recommendations to receive booster).
- 16. Has received or plans to receive immunoglobulins or any blood or blood products within 90 days before study vaccination and throughout the study.
- 17. Reports chronic use (more than 14 continuous days) of any medication that may be associated with changes in immune function including, but not limited to, systemic corticosteroids exceeding 20 mg/day of prednisone equivalent, allergy injections, immunoglobulins, interferons, immunomodulators, cytotoxic drugs, or other similar or toxic drugs within 6 months of study vaccination. Note: The use of low-dose topical, ophthalmic, inhaled, intra-articular and intranasal steroid preparations is permitted.

#### 5.2.3. Other exclusions

- 18. Pregnant or lactating female.
- 19. Female participant planning to become pregnant or planning to discontinue contraceptive precautions within 1 month following study vaccination.
- 20. Participant is an employee or family member of the investigator or study site personnel.

#### 5.3. Screen failures

A screen failure is an individual who consents to participate in this study but is not entered in the study/assigned to a study intervention.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Limited data for screening failures (including informed consent, inclusion/exclusion criteria, demographic data, pregnancy reason for screening failure and any SAEs that occurred at the visit) will be collected and reported in the eCRF.

If the investigator believes there is a reasonable justification to do so, all screening procedures may be repeated (maximum 1 re-screening per participant is allowed) under a new participant number. The participant can only be randomized into the study once the investigator receives the results and confirms the eligibility criteria.

Participants with hematological/biochemical values out of normal range which are expected to be temporary may be re-screened at a later date, as per the above conditions.

# 5.4. Criteria for temporarily delaying enrollment, randomization and study intervention administration

Enrollment, randomization and study intervention administration may be postponed within the 14-day screening interval until transient conditions cited below are resolved:

- Acute disease and/or fever at the time of enrollment and/or study intervention administration. Refer to the Section 1.3 for definition of fever and oral temperature in this study.
- Participants with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may be enrolled and/or dosed at the discretion of the investigator.
- If antipyretics and/or analgesics and/or antibiotics have been used within 3 days prior to study intervention administration.

#### 6. STUDY INTERVENTION AND CONCOMITANT THERAPY

Refer to the Definition of terms for the definition of study intervention.

# 6.1. Study interventions administered

Refer to Section 1.2 for the study intervention administration schedule. Table 6 and Table 7 describe study interventions to be administered for Part A and Part B, respectively.

Table 6 Part A study interventions administered

| | mRNA-CR-04 | | Placebo |
|---|---|---|---|
| Study intervention#:<br>Group 1 | COV08A/DL001Z | | PL001Z |
| Group 2 | COV08B/DL001Z | PL001Z | |
| Group 3 | COV08C | | PL001Z |
| Study intervention formulation#:<br>Group 1 | GSKVx000000037755 (Dose Aa GSKVx000000037754);<br>Excipients; Water for injections | | |
| Group 2 | GSKVx000000037755 (Dose Ab GSKVx000000037754);<br>Excipients; Water for injections | GSKVx000000037755 (Dose Ab GSKVx000000037754); Excipients; Water for | |
| Group 3 | GSKVx000000037755 (Dose Ac GSKVx000000037754);<br>injections | GSKVx000000037755 (Dose Ac GSKVx000000037754); Excipients; Water for | |
| Presentation:<br>Group 1 | Concentrate for dispersion for injection (vial) Solution for dispersion for injection (vial) | | Solution for injection (vial) |
| Group 2 | Concentrate for dispersion for injection (vial) Solution for dispersion for injection (vial) | | Solution for injection (vial) |
| Group 3 | Dispersion for injection (vial) | | Solution for injection (vial) |
| Type: | Investigational | | Placebo |
| Product category: | Biologic | | Drug |
| Route of administration: | IM | | IM |
| Location | Deltoid | | Deltoid |
| Directionality | NA | | NA |
| Laterality* | Non-Dominant | Non-Dominant | |
| Number of doses to be administered | 1 | 1 | |
| Volume to be administered by dose ** | 0.3 mL | 0.3 mL | |
| Packaging and labeling: | Refer to the PM for more details | | Refer to the PM for more details |
| Manufacturer: | GSK | | Hospira |

43 07 Feb 2024

Ab: Antibody; IM: Intramuscular; GSK: GlaxoSmithKline Biologicals SA; NA: Not applicable; PM: Pharmacy manual.

\*The non-dominant arm is the preferred arm of injection. In case it is not possible to administer the study intervention in the non-dominant arm, an injection in the dominant arm may be performed.

<sup>\*\*</sup>Refer to the PM for the volume after reconstitution.

<sup>#</sup>Coding serves for internal sponsor anonymization

Table 7 Part B study interventions administered

| | | mRNA-CR-04 | | | |
|---|---|---|---|---|---|
| Study Groups | Part B 3 µg | | Part B 10 µg | Part B Placebo | |
| Study intervention <sup>#</sup> | COV08D/DL001Z | | COV08A/DL001Z | | PL001Z |
| Study intervention formulation#: | GSKVx000000037755 (Dose Ad GSKVx000000037754); Excipients; Water for injections injections | | GSKVx000000037755 (Dose Aa<br>GSKVx000000037754); Excipients;<br>Water for injections | Excipients;<br>Water for<br>injections | Excipients; Water for injections |
| Presentation: | Concentrate for dispersion for injection (vial) | Solution for dispersion for injection (vial) | Concentrate for dispersion for injection (vial) | Solution for dispersion for injection (vial) | Solution for injection (vial) |
| Type: | Investigational | | Investigational | Placebo | |
| Product category: | | Biol | ogic | | Drug |
| Route of administration: | | Į. | M | | IM |
| Location | | Del | Itoid | | Deltoid |
| Directionality | | N | IA | | NA |
| Laterality* | | Non-Do | ominant | | Non-Dominant |
| Number of doses to be<br>administered | 1 | | | | 1 |
| Volume to be administered by dose ** | 0.3 mL | | | | 0.3 mL |
| Packaging and labeling: | Refer to the PM for more details | | | | Refer to the PM for more details |
| Manufacturer: | | G | SK | | Hospira |

Ab: Antibody; IM: Intramuscular; GSK: GlaxoSmithKline Biologicals SA; NA: Not applicable; PM: Pharmacy manual.

<sup>\*</sup>The non-dominant arm is the preferred arm of injection. In case it is not possible to administer the study intervention in the non-dominant arm, an injection in the dominant arm may be performed.

<sup>\*\*</sup>Refer to the PM for the volume after reconstitution.

<sup>#</sup>Coding serves for internal sponsor anonymization

## 6.2. Preparation, handling, storage, and accountability

The study interventions must be stored in a secured place within the temperature range specified on the study intervention's label. The storage temperature should be continuously monitored and recorded with a calibrated (if not validated) temperature monitoring device.

Only unblinded staff should be allowed access to the study interventions. Storage conditions will be assessed by a sponsor study contact during pre-study activities. Refer to the PM for more details on storage and handling of the study interventions.

## 6.3. Measures to minimize bias: randomization and blinding

This is a dose-escalation, observer-blind, randomized study.

## 6.3.1. Participant identification

Participant identification numbers will be assigned sequentially to the individuals who have consented to participate in the study by using an automated internet-based system (e.g., IRT).

## 6.3.2. Randomization to study intervention

The randomization of study interventions will be performed using the IRT system.

## 6.3.3. Intervention allocation to the participant

In Part A of the study, approximately 72 participants will be enrolled with 24 participants per group. These 24 eligible participants will be randomly assigned to investigational mRNA-CR-04 vaccine or saline placebo in a (3:1) ratio. In Part B of the study, approximately 42 participants will be enrolled and randomly assigned to 3  $\mu$ g investigational mRNA-CR-04 vaccine, 10  $\mu$ g investigational mRNA-CR-04 vaccine, or saline placebo in a (3:3:1) ratio.

## 6.3.4. Blinding and unblinding

In Part A of the study, data will be collected in an observer-blind manner. The participant, the site and sponsor personnel involved in the clinical evaluation of the participants are blinded while other study personnel may be aware of the treatment assignment. To do so, study interventions will be prepared and administered by qualified study personnel who will not participate in data collection, evaluation, review, or the entry of any study endpoint data (i.e., reactogenicity, safety, immunogenicity). In Part B of the study (i.e., following the Part A Day 15 interim analysis), continuation of the observer-blind design will be restricted to study participants and site personnel involved in the clinical evaluation of the participants, while sponsor personnel will no longer remain blinded to treatment assignment.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Unblinding a participant's individual study randomization number should occur ONLY in case of a medical emergency when this information is essential for the clinical management or welfare of the participant.

In case of emergency, the investigator can have unrestricted, immediate and direct access to the participant's study intervention information via the IRT. The investigator may contact Signant Health support (refer to Table 8) if help is needed to access participant's study intervention information (i.e., if the investigator is unable to access IRT).

A physician other than the investigator (e.g., an emergency room physician) or participant may also request emergency access to the participant's study intervention information via the investigator.

## Table 8 Contact information for emergency unblinding

#### Signant Health support

Available 24/24 hours and 7/7 days

The Signant Health support is available by phone and email

US: 1-888-794-0122

IRTHelpdesk@SignantHealth.com

A participant may continue in the study if that participant's treatment assignment is unblinded.

GSK's Global Safety staff may unblind the intervention assignment for any participant with an SAE. If the SAE requires that an expedited regulatory report be sent to one or more regulatory agencies, a copy of the report, identifying the participant's intervention assignment, may be sent to investigators in accordance with local regulations and/or GSK policy.

# 6.4. Study intervention compliance

When the study intervention is administered at the site, participants will receive the dose of study vaccine directly from the investigator or designee, under medical supervision. The date and time of administration of each study intervention dose in the clinic will be recorded in the source documents.

#### 6.5. Dose modification

Not applicable.

# 6.6. Continued access to study intervention after the end of the study

Not applicable.

#### 6.7. Treatment of overdose

An overdose is any dose of study vaccine given to a participant that exceeds the planned dose for an individual participant within a given group.

There is no specific treatment recommended for an overdose.

Any overdose must be promptly reported to the CRO team within 24 hours. Overdose itself is not to be reported as an AE. However, any AEs associated with the overdose are to be reported in the relevant AE/SAE sections of the eCRF.

In the event of an overdose, the investigator should:

- 1. Contact the CRO medical monitor immediately.
- 2. Closely monitor the participant for any AE/SAE and laboratory abnormalities for at least 3 days. Refer the participant to a higher level of care as clinically indicated.
- 3. Document the quantity of the excess dose in the eCRF.

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the medical monitor based on the clinical evaluation of the participant.

## 6.8. Concomitant therapy

At each study visit/contact, the investigator(s) or their delegate(s) should question the participant about all medications/products taken, and vaccinations received by the participant.

The following concomitant medication(s)/product(s)/vaccine(s) must be recorded in the eCRF:

- All concomitant medications, except vitamins and dietary supplements, administered during the entire study.
- Any concomitant use of antipyretic/analgesic medication from Day 1 to Day 7 after vaccination.
- Any concomitant vaccination administered in the period starting 30 days before study intervention administration and ending 30 days after vaccination.
- Any booster COVID-19 vaccines received during the study will be recorded.
- All concomitant medication associated with an AE, including vaccines/products, administered after study intervention vaccination (Day 1 to Day 31).
- All concomitant medication leading to discontinuation of the study intervention or elimination from the analysis, including products/vaccines. Please refer to Section 5.2.2 and Section 9.3.1 for further details.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

• All concomitant medication which may explain/cause/be used to treat an SAE/AESI including vaccines/products, as defined in Section 8.4.1. These must also be recorded in the electronic AE report.

The medical monitor should be contacted if there are any questions regarding concomitant or prior therapy.

# 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

# 7.1. Discontinuation of study intervention

Not applicable.

# 7.1.1. Contraindications to subsequent study interventions administration

Not applicable.

## 7.2. Participant discontinuation/withdrawal from the study

Individual participants may withdraw from the study at any time at their own request for any reason without prejudice to their future medical care by the investigator or at the study site.

A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for them since the date of withdrawal/last contact.

From an analysis perspective, a study 'withdrawal' refers to any participant who did not return for the concluding visit planned in the protocol.

Investigators will attempt to contact participants who do not return for scheduled visits or follow-up.

At the time of discontinuing from the study, if possible, an early termination visit should be conducted, as shown in the SoA (Section 1.3). See SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.

All data and samples collected up to and including the date of withdrawal of/last contact with the participant will be included in the study analyses.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

The primary reason for study withdrawal will be documented in the eCRF based on the list below:

| Reasons | Additional items/Sub-reasons |
|---|---|
| AE | Unsolicited AE<br>Solicited AE |
| Lost to follow-up | Participant Relocated Other, specify Unknown |
| Study Terminated by Sponsor | |
| Withdrawal by Participant (not due to an AE) | Participant Relocated Other, specify |
| Other | Specify |

AE: Adverse event

Participants who are withdrawn from the study because of AEs/SAEs must be clearly distinguished from participants who are withdrawn for other reasons. Investigator will follow participants who are withdrawn from the study due to an AE/SAE until the event is resolved (see Section 10.3.5.5).

## 7.3. Lost to follow-up

Participants will be considered 'lost to follow-up' if they fail to return for scheduled visits and cannot be contacted by the study site.

Please refer to the PM for a description of actions to be taken before considering the participant lost to follow-up.

## 8. STUDY ASSESSMENTS AND PROCEDURES

Protocol waivers or exemptions are only permitted when necessary for the management of immediate safety concerns for the participant.

Immediate safety concerns should be discussed with the CRO team as soon as they occur or when the study team becomes aware of them. The purpose of this communication is to determine if the participant(s) should discontinue the study intervention.

Study procedures and their timing are summarized in the SoA (Section 1.3).

All screening evaluations must be completed, and the results reviewed before confirming that potential participants meet all eligibility criteria.

The investigator will maintain a log of all participants screened. All relevant information, such as confirmation of eligibility and reasons for screening failure will be mentioned in this screening log.

Procedures conducted as part of routine clinical management (e.g., hematologic profiles), and obtained before the participant signed the ICF, may be used for screening and/or for

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

establishing a clinical baseline (provided the procedure met protocol specified criteria and was performed within the time frame defined in the SoA in Section 1.3).

The PM provides the investigator and site personnel with detailed administrative and technical information that does not impact participant safety.

During special circumstances (e.g., COVID-19 pandemic), certain study procedures may be adapted to protect the participant's welfare, and as far as possible to ensure the potential benefit to the participant and promote data integrity. See Section 8.10.

## 8.1. Administrative procedures

All screening procedures, except the SARS-CoV-2 PCR test, need to be performed within 14 days of Visit 1 (see Section 5.1). A SARS-CoV-2 PCR test needs to be performed within 7 days of Visit 1. A sample may be collected for repeat testing at any time (but only once to assess eligibility) before Visit 1.

## 8.1.1. Collection of demographic data

At screening, record demographic data such as year of birth, sex, race, and ethnicity in the participant's eCRF.

Collection of sex, race and ethnicity data is necessary to assess and monitor the diversity of the trial participants, and to determine if the trial participants are truly representative of the impacted population.

### 8.1.2. Medical/vaccination history

At screening, obtain the participant's medical/vaccination history by interviewing the participant and/or review of the participant's medical records. Record any pre-existing conditions, vaccination history, signs and/or symptoms present prior to study intervention in the eCRF.

## 8.1.3. Distribution of eDiary or installing the application for devices

Participants will be encouraged to bring their own devices at screening visit, or if not feasible, at Visit 1 (Day 1). The study staff will check the compatibility of participant's device (e.g., smart phone or tablet) with respect to eDiary application.

At Visit 1 (Day 1), participant will download the eDiary application on his/her own electronic device or will receive an electronic device to record information related to his/her health and participation in the study. The participant will also be trained on the use of eDiary.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Refer to Section 8.4.1 for details of collection of safety information and Section 10.3.5 for guidelines.

For the vendors that will perform eDiary-related activities, please refer to the separate list of vendors.

# 8.2. Immunogenicity assessments

Blood samples will be taken to assess both the humoral and cellular immune responses induced by the vaccine candidate on Day 1, Day 15, Day 31, and Month 6.

In addition, biological samples will be used for research planned in the protocol and for purposes related to the improvement, development and quality assurance of the laboratory tests described in this protocol.

Findings in this or future studies may make it desirable to use samples acquired in this study for research not planned in this protocol. In this case, all participants in countries where this is allowed will be asked to give consent to allow GSK or a contracted partner, to use the samples for further research. The further research will be subject to prior IEC/IRB approval, if required by local legislation.

Information on further research and its rationale can be obtained from GSK.

Sample testing will be done in accordance with the recorded consent of the individual participant.

By default, collected samples will be stored for a maximum of 20 years. This storage period begins when the last participant performs the last study visit. This timeline can be adapted based on local laws, regulations or guidelines requiring different timeframes or procedures. In all cases, the storage period should be aligned with participant's consent. These additional requirements must be formally communicated to, discussed, and agreed with GSK.

### 8.2.1. Biological samples

Table 9 Biological samples

| Sample type | Quantity | Unit | Timepoint | Subset name |
|---|---|---|---|---|
| | | | Screening (D-7 to D-1) | All screened participants |
| Nasopharyngeal swab for | NA | NIA | Visit 1 (D1) | |
| SARS-CoV-2 test | INA | NA | Visit 2 (D8) All enrolled participants | |
| | | | Visit 3 (D15) | |
| Blood for FSH | ~2.5 | mL | Screening (D-14 to D-1) | Female participants to confirm non-childbearing potential |
| Blood for Troponin I | ~2.5 | mL | Screening (D-14 to D-1) | All screened participants |
| Blood for Troponiiri | ~2.5 | IIIL | Visit 2 (D8) | All enrolled participants |
| | | mL | Screening (D-14 to D-1) | All screened participants |
| Blood for hematology/ | ~6 | | Visit 1 (D1) | |
| biochemistry | | | Visit 2 (D8) | All enrolled participants |
| | | | Visit 3 (D15) | |
| Blood (serum) for vaccine- | | | Visit 1 (D1) | |
| induced humoral immune | ~15 | mL | Visit 3 (D15) | All enrolled participants |
| response and to assess SARS- | 10 | IIIL | Visit 4 (D31) | All chroned participants |
| CoV2 N protein serology | | | Visit 5 (M6) | |
| | | | Visit 1 (D1) | |
| Blood (PBMCs) for cellular | ~50 | l mL | Visit 3 (D15) | All enrolled participants |
| immune response | 30 | Visit 4 (D31) | 7 til omonou participanto | |
| D. D. 5011 5 111 11 11 11 11 | | | Visit 5 (M6) | |

D: Day; FSH: Follicle stimulating hormone; M: Month; N: Nucleocapsid; NA: Not applicable; PBMC: Peripheral blood mononuclear cell.

## 8.2.2. Laboratory assays

Following laboratory assays will be performed (Table 10).

- PCR assay will be used to detect SARS-CoV-2 infection. If the sample is positive and sufficient material is available, sequencing of the SARS-CoV-2 isolate will be performed by genomic RNASeq.
- Serological assay to monitor the asymptomatic infection will be performed using an ECL to measure serum-binding Abs IgG levels specific for N protein of SARS-CoV-
- The vaccine-induced humoral immunity will be evaluated using serological assays determining the capacity of the serum of SARS-CoV-2 vaccinated participants to neutralize pseudoviruses bearing S protein from vaccine encoded SARS-COV-2 and from the WT (D614G).
- Further characterization of the humoral immune response will be performed using ECL for measurement of IgG antibodies binding to the SARS-CoV-2 S protein (at least vaccine encoded SARS-CoV-2 variant and WT).
- The cell-mediated immunity will be evaluated by assessing the frequency of SARS-CoV-2 S-specific CD4+ and CD8+ T-cells expressing specific activation or immune markers using ICS per million of total CD4+ or CD8+ T-cells respectively.

## Table 10 Laboratory assays

| Assay Type | System | Component | Challenge | Method | Laboratory** |
|---|---|---|---|---|---|
| Humoral immunity | Serum | Anti-S binding IgG<br>Ab | | | PPD |
| (antibody<br>determination)* | Serum | Anti-SARS-CoV-2 neutralizing titer | IVA | Pseudo<br>Neutralization<br>assay | Nexelis |
| Cell-mediated immunity | PBMCs | CD4+/CD8+ T-cells<br>expressing IL-<br>2/IFNγ/TNFα/IL-<br>13/IL-17/4-<br>1BB/CD40L | Peptide pools<br>covering the<br>SARS-CoV-2<br>S protein | ICS | GSK |
| Detection of SARS-<br>CoV-2 Infection | Serum | Anti-N IgG Ab | NA | ECL | PPD |
| Detection of SARS-<br>CoV-2 Infection | Nasopharyngeal<br>Swab | SARS-CoV-2 RNA | NA | RT-PCR | PPD |
| Sequencing of<br>SARS-CoV-2<br>Isolates | Nasopharyngeal<br>Swab | SARS-CoV-2 RNA | NA | RNASeq | PPD |

Ab: Antibody; CD40L: Cluster of differentiation 40 ligand; 4-1BB: CD137 (tumor necrosis factor receptor superfamily 9); CRO: Contract research organization; ECL: Electro-chemiluminescence assay; GSK: GlaxoSmithKline Biologicals SA; ICS: Intracellular cytokine staining; IgG: Immunoglobulin G; IFNy: Interferon gamma; IL-2: Interleukin-2; IL-13: Interleukin-17; NA: Not applicable; N: Nucleocapsid; PPD: Pharmaceutical Product Development; RNASeq: RNA Sequencing; RT-PCR: Real-time polymerase chain reaction; S: Spike; TNFα: Tumor necrosis factor alpha; WT: Wild type.

Please refer to Section 10.2 for further details.

The addresses of clinical laboratories used for sample analysis are provided in a separate document accompanying this study protocol.

GSK clinical laboratories have established a quality system supported by procedures. The activities of GSK clinical laboratories are audited regularly for quality assessment by an internal (sponsor-dependent) but laboratory-independent quality department.

53

<sup>\*</sup> Measurement of humoral immunity against vaccine encoded SARS-CoV-2 and WT strains.

<sup>\*\*</sup> Refer to the list of clinical laboratories for details.

### 8.2.3. Immunological read-outs

Table 11 Immunological read-outs

| Blood san | pling timepoint | Subset name | No. participants | Component |
|---|---|---|---|---|
| Type of contact<br>and timepoint | Sampling timepoint | | | |
| Visit 1 (D1) | Pre-Dose 1 | All enrolled participants | 72 (Part A) +<br>42 (Part B) | SARS-CoV-2 neutralizing titer Anti-S binding IgG Ab Anti-N IgG Ab S-specific CD4+/CD8+ T-cells |
| Visit 3 (D15) | 14 days Post-Dose 1 | All enrolled participants | 72 (Part A) +<br>42 (Part B) | SARS-CoV-2 neutralizing titer Anti-S binding IgG Ab Anti-N IgG Ab S-specific CD4+/CD8+ T-cells |
| Visit 4 (D31) | 30 days Post-Dose 1 | All enrolled participants | 72 (Part A) +<br>42 (Part B) | SARS-CoV-2 neutralizing titer Anti-S binding IgG Ab Anti-N IgG Ab S-specific CD4+/CD8+ T-cells |
| Visit 5 (M6) | 6 months Post-Dose 1 | All enrolled participants | 72 (Part A) +<br>42 (Part B) | Anti-SARS-CoV-2 neutralizing titer Anti-S IgG Ab Anti-N IgG Ab S-specific CD4+/CD8+ T-cells |

Ab: Antibody; D: Day; IgG: Immunoglobulin G; M: Month; N: Nucleocapsid; S: Spike.

## 8.2.4. Cytology

Not applicable.

# 8.2.5. Immunological correlates of protection

No validated mechanistic immunological correlate of protection has been demonstrated so far for the antigens used in the study intervention.

# 8.3. Safety assessments

Planned timepoints for all safety assessments are provided in the SoA (Section 1.3).

## 8.3.1. Physical examination

• At screening and prior to dosing at Visit 1 (Day 1), the investigator will perform a physical examination of the participant. The following information needs to be recorded in the eCRF: weight, oral temperature, resting vital signs (before blood collection for laboratory test); systolic/diastolic blood pressure and heart rate after at least 10 minutes of rest. If the participant reported any pre-existing medical condition, the investigator would extend the physical examination according to his/her medical judgment to ensure that the participant meets all the eligibility criteria. Height and BMI will only be recorded at screening.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- A targeted physical examination at each study visit after the Screening visit, will be performed only if the participant indicates during questioning that there might be some underlying pathology(ies) or if deemed necessary by the investigator or delegate.
- If the investigator determines that the participant's health on the day of study intervention administration temporarily precludes dosing, the visit will be rescheduled. Refer to the Section 5.4 for the list of criteria for temporary delay of study intervention administration.
- Treatment of any abnormality observed during post-vaccination visits must be performed according to local medical practice outside this study or by referral to an appropriate health care provider and recorded as AE.

## 8.3.2. Pre-dosing body temperature

The body temperature of each participant needs to be measured orally prior to the study vaccine administration and recorded in the eCRF. If the participant has fever on the day of dosing, the study intervention administration visit will be rescheduled. Refer to the SoA (Section 1.3) for the definition of fever for this study and preferred location for body temperature measurement.

## 8.3.3. Pregnancy test

Female participants of childbearing potential must perform a urine pregnancy test before the administration of the study intervention. At screening, if time allows, a serum pregnancy test can be done, in place of the urine pregnancy test, as per local requirements. Pregnancy testing must be done even if the participant is menstruating at the time of the study visit. The study intervention may only be administered if the pregnancy test is negative.

Refer to Section 8.4.6 for the information on study continuation for participants who become pregnant during the study.

For WONCBP, document the specific reason for not performing a pregnancy test in the eCRF.

#### 8.3.4. EKGs

• 12-lead EKGs will be obtained as outlined in the SoA (see Section 1.3) using an EKG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.

## 8.3.5. Warnings and precautions to administration of study intervention

Vital signs, including oral temperature, systolic/diastolic blood pressure and heart rate after at least 10 minutes of rest for each participant needs to be measured prior to administration of study intervention, i.e., at Visit 1. Collected information will be recorded in the eCRF.

## 8.3.6. Clinical safety laboratory tests

- See Section 10.2.1 for the list of clinical laboratory tests to be performed in accordance with lab manual and the SoA (Section 1.3).
- The investigator must review the laboratory results, document this review, and record any clinically significant changes occurring during the study as an AE. The laboratory results must be retained with source documents.
- Abnormal laboratory findings associated with the underlying disease are not considered clinically significant unless judged by the investigator to be more severe than expected for the participant's condition.
- All laboratory tests with values considered clinically significantly abnormal during participation in the study or within 31 days after the last dose of study intervention should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the investigator or medical monitor.
  - In the absence of a diagnosis, abnormal laboratory findings assessments or other abnormal results the investigator considers clinically significant will be recorded as an AE or SAE, if they meet the definition of an AE or SAE (refer to Section 10.3.1 and Section 10.3.2).
  - If clinically significant values do not return to normal/baseline within a period of time judged reasonable by the investigator, the etiology should be identified, and the sponsor notified.
  - If laboratory values from non-protocol-specified laboratory tests performed at the institution's local laboratory require a change in participant management or are considered clinically significant by the investigator (e.g., SAE or AE), then the results must be recorded.
- Analyses of safety laboratory samples collected at Day 1 through the EoS will be performed at the central laboratory using the same grading standards.
- Laboratory data will be graded according to the FDA guidance for industry "Toxicity grading scale for healthy adults and adolescent volunteers enrolled in preventive vaccine clinical trials" dated September 2007 [FDA, 2007]. These laboratory values serve as guidelines and are dependent upon laboratory normal parameters. Normal reference ranges should be provided to demonstrate that they are appropriate. Any laboratory parameters not listed in Table 19 and Table 20 (Section 10.2.2) will not be graded and will be assessed on case-by-case basis.

## 8.3.7. Study holding rules and safety monitoring

Safety monitoring is specified in the SoA (Section 1.3), Section 8.3.7.1 and Table 12.

For the vendors that will perform safety monitoring activities, please refer to the separate list of vendors.

#### 8.3.7.1. Staggered administration of study intervention

Part A of the study will be conducted in a staggered manner to ensure maximum safety of the participating participants.

- Within each group, 8 sentinel participants (6 receiving the mRNA-CR-04 vaccine and 2 receiving the placebo) will first be enrolled and vaccinated.
- Enrollment of participants in Group 1 and Group 2 will be done in parallel with the first participant to be enrolled in Group 1. The first and second sentinel participant in each group will be vaccinated and followed-up for 24 hours before the next sentinel participant can be vaccinated. If no safety concerns are identified (as confirmed through individual phone call TC1, see Table 1), vaccination of the remaining sentinel participants in the same group will then continue with an interval of at least 60 minutes between participants. Additionally, an interval of at least 60 minutes will be maintained between the vaccination of sentinel participants across groups.
- If no safety concerns are identified by the iSRC during the review of unblinded Day 8 safety data of sentinel participants from Group 1 and Group 2, the remaining participants in these groups may receive the study intervention without limitation of the number of participants per day or the time between consecutive participants. Additionally, vaccination of sentinel participants in Group 3 may be initiated.
- If no safety concerns are identified by the iSRC review of unblinded Day 8 safety data of sentinel participants from Group 3, the remaining participants in Group 3 may receive the study intervention without limitation of the number of participants per day or the time between consecutive participants.

All participants will be closely observed (visibly followed, no specific procedure) during the 60 minutes after dose administration.

In addition to iSRC, blinded data will be reviewed by the SRT. The SRT and iSRC will meet regularly to review safety data throughout the study and may request escalation to the GSB to address any potential safety concerns or study holds at any point during the study. See Section 8.3.7.3.

In Part B of the study, irrespective of dose, all participants will be enrolled in parallel, and the SRT will also be able to review unblinded data.

#### 8.3.7.2. Outcome of safety evaluation

Outcome of safety evaluations will be documented and provided in a written way to the investigator. Refer to iSRC charter for more details.

- If **no safety** signal is observed, the favorable outcome of the safety evaluations by the iSRC will be documented and provided, authorizing the investigator to start the enrollment and study intervention administration to the remaining participants in the group and the sentinel participants in the next group.
- If a safety signal is observed during the safety evaluations or if any of the holding rules is met, the iSRC Chair is responsible for the urgent communication and escalation of the concern to the GSB. The GSB will decide and communicate whether to suspend, modify or continue the conduct of the study on all groups or on selected groups, including the rationale for the decision to put the study intervention administration on hold or not.
- The study sponsor will be accountable for notifying the decision whether to suspend, modify or continue the conduct of the study on all groups or on selected groups to the CRO. The CRO will be responsible to inform all investigators of this decision.

## 8.3.7.3. Study holding rules

The safety holding rules are defined in the Table 12. Holding rules 1a-d will be assessed by the investigator on a continuous basis. Meeting any of these holding rules will trigger a hold of study intervention administration irrespective of number of participants enrolled and/or timing of the event. Holding rules 2a-c will be assessed by the iSRC during the safety evaluations on unblinded data.

These holding rules have been written under the assumption that the safety data from all participants will be available. If the data from all participants are not available (i.e., in case a participant is lost to follow-up), then the holding rules will be assessed on a prorata basis (expressed as percentage of participants to be evaluated) i.e., 3 out of 6 sentinel participants or 30% of all participants, whichever is met earlier.

Of note, no formal holding rules will be applied for other safety data such as non-life-threatening SAEs, missed visits due to study intervention related AEs, Grade 1 and Grade 2 solicited and unsolicited AEs in the 7-day follow-up period (Day 1 to Day 7) and unsolicited AEs collected from Day 8 to Day 31 after study intervention administration. However, if available, these data will also be reviewed by the iSRC to allow an overall assessment of the benefit/risk ratio of study intervention administration.

## Table 12 Study holding rules

| Holding rule | Event (per dose and per individual study group) | Number of participants<br>to pause vaccination in<br>all groups, pending<br>further evaluation by<br>iSRC |
|---|---|---|
| 1a | Death or any life-threatening SAE regardless of causality | ≥1 |
| 1b | Any non-life-threatening SAE that cannot be reasonably attributed to a cause other than vaccination as per investigator or sponsor assessment | ≥1 |
| 1c | Any withdrawal from the study (by investigator or participant request) following a Grade 3 AE | ≥1 |
| 1d | Any administration site or systemic solicited AE leading to hospitalization, OR Necrosis at the injection site, Each with an event onset within the 7-day (Day 1-7) post-vaccination period | ≥1 |
| 2a* | Any Grade 3 solicited administration site events, with an event onset within the 7-day (Day 1-7) post-vaccination period | ≥3/6 or 30%** |
| 2b* | Any Grade 3 solicited systemic events, with an event onset within the 7-day (Day 1-7) post-vaccination period | ≥3/6 or 30%** |
| 2c* | Any Grade 3 unsolicited AE, that can be reasonably attributed to the vaccination as per investigator or sponsor assessment, with an event onset within the 7-day (Day 1-7) post-vaccination period OR Any Grade 3 or above abnormality in pre-specified hematological or biochemical laboratory parameters with an event onset within the 8-day (Day 1-8) post-vaccination period except for non-clinically significant leukopenia | ≥2/6 or 10%*** |

AE: Adverse event; iSRC: Internal safety review committee; SAE: Serious adverse event.

Rule 2a-2c will be analyzed and reviewed during the scheduled iSRC meetings. During these scheduled iSRC meetings, iSRC will decide to:

- allow for dosing of the remaining non-sentinel participants (12 receiving mRNA-CR-04 and 4 receiving placebo) within the same group
- allow for randomization of the sentinel participants in the next group.

More details on the composition, objectives, and responsibilities of the iSRC, and the schedule and conduct of the iSRC meetings will be described in the iSRC charter.

59

<sup>\*</sup>Refer to the FDA guidance for industry "Toxicity grading scale for healthy adults and adolescent volunteers enrolled in preventive vaccine clinical trials" [FDA, 2007]. Any laboratory parameters not listed in Section 10.2.2 will not be graded and will be assessed on case-by-case basis.

<sup>\*\*3/6</sup> sentinel participants or 30% of all participants, whichever is met earlier.

<sup>\*\*\*2/6</sup> sentinel participants or 10% of all participants, whichever is met earlier.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

If a holding rule is met, the investigator must suspend enrollment and administration of the study intervention and inform the CRO team immediately (holding rules 1a-d). Refer to Table 16 for contact information.

The CRO team will inform the investigator if holding rules 2a-c are met. Investigators will be responsible to inform the IRB/IEC if a holding rule has been met.

The following communication sequence must be followed when a holding rule 1a-1d is met:

- The concerned site staff must put study intervention randomization and administration on hold.
- The concerned site staff must immediately inform the CRO team contact defined in the Section 8.4.6.
- Enrollment and intervention allocation through IRT will be stopped on a study level.
- The CRO team will inform all investigators about the stopping of enrollment and intervention.
- All informed site staff will confirm to the CRO team that action has been taken providing appropriate documentation to the CRO team.
- The CRO team will inform GSK and provide the blinded data to GSK's CSL for further SRT and GSK GSB review.
- The CRO team will forward the relevant unblinded safety information to iSRC for evaluation.
- Based on the recommendation from iSRC, GSK's GSB will make the decision whether the study can resume, be modified, or stopped. GSK will notify the CRO team on this decision. The CRO team will notify all investigators on this decision.
- Depending on the outcome of the safety evaluation, the study will be re-started, terminated, or resumed under a protocol amendment.

The following communication sequence must be followed when a holding rule 2a-2c is being met:

- The study CSL will ensure that the CRO team is notified upon meeting holding rules 2a-2c.
- The CRO team will inform all the sites that a holding rule is met. Following this notification, the study intervention administration should be put on hold.
- All informed site staff will confirm to the CRO team that action has been taken providing appropriate documentation to the CRO team.
- GSK will further evaluate the case with the iSRC and GSK GSB and will take the decision to stop or to restart the study intervention administration or to amend the protocol. GSK will notify the CRO team on this decision and the CRO team will inform all site staff.

#### Risk assessment:

- Figure 2 illustrates that with 6 participants receiving the mRNA-CR-04 vaccine per group:
  - Rule 1: when at least 1 SAE is observed within 6 participants receiving the mRNA-CR-04 vaccine, there is 90% probability of not holding for a 1.7% SAE true incidence and 80% (=1-20%) probability of holding it for an SAE true incidence >23%.
  - Rule 2a-2b: when at least 3 participants with an AE are observed within 6 participants receiving the mRNA-CR-04 vaccine, there is 90% probability of not holding for a 20% AE true incidence and 80% (=1-20%) probability of holding it with a true AE incidence >58%.
  - Rule 2c: when at least 2 participants with an AE are observed within 6 participants receiving the mRNA-CR-04 vaccine, there is 90% probability of not holding for a 9% AE true incidence and 80% (=1-20%) probability of holding it with a true AE incidence >42%.
  - With 18 participants receiving the mRNA-CR-04 vaccine, and rule 1 (1/18), there is 90% probability of not holding for a 0.59% AE true incidence and 80% (=1-20%) probability of holding it with a true incidence >8.5%.

Figure 2 Probability of not meeting holding rules 1 and 2 for 8 participants per study group



#### 8.3.7.4. SRT and iSRC evaluation

The study will be overseen by an iSRC operating under a charter. Core members of the iSRC will include a GSK safety physician, a CSL and a biostatistician who are not otherwise involved in the conduct of the project. The iSRC safety reviews will be conducted using unblinded data. The iSRC will have access to the participant randomization and will review unblinded data.

In addition to the iSRC, the project SRT will review blinded data until the Part A Day 15 interim analysis, and unblinded data subsequently, on a regular basis throughout the study.

The iSRC will review accumulated unblinded safety data of the sentinel participants of each group up to 7 days post-vaccination. The iSRC will include all safety data sources in their Day 8 safety review (i.e., solicited safety data, unsolicited safety data, SAEs and AESIs, as well as laboratory safety data). If no pre-defined holding rule is met (refer to Section 8.3.7.3) or if no safety signal is observed the remaining participants in the group can be vaccinated and vaccination in the next group can be initiated.

In case the iSRC, through the in-stream data monitoring of all the accumulated safety data available detects that a holding rule is met, the study vaccination will be temporarily paused in all study groups and sites pending review of safety data by the iSRC. The iSRC will make relevant recommendations to the GSB chair(s), who will make the final decision whether vaccination can be safely resumed or not.

In addition, at any time during the study, if one of the holding rules 1a through 1d (refer to Table 12 for details) is met, the investigator will immediately inform the CRO team. Vaccination will be paused and an urgent ad-hoc meeting of the iSRC will be called to thoroughly review the event(s) and recommend to the GSB whether vaccination can be safely resumed or not. The GSB chair(s) will make the final decision whether vaccination can be safely resumed or not.

In Part B of the study, the iSRC will only be requested to review unblinded data if a study holding rule is met or if the SRT identifies a safety concern through in-stream data monitoring of unblinded data.

#### 8.3.8. Cardiac adjudication

Myocarditis and pericarditis are considered as important potential risk and are collected as AESI. All surveillance EKGs occurring at Screening, Day 8, and unscheduled visits, will be reviewed by an independent external cardiologist in a blinded fashion to identify potential myocarditis or pericarditis cases. All EKGs identified with changes suggestive of potential myocarditis and pericarditis and related available medical records requested from treating cardiologists evaluating potential cases of myocarditis and pericarditis, will then be provided to an independent external adjudication committee for case adjudication according to the case definition from the Brighton Collaboration [Sexson, 2022]. The committee members will remain blinded to study intervention assignment.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

For details on who will perform the reading and adjudication activities, please refer to the separate list of vendors.

## 8.4. AEs, SAEs, and other safety reporting

For definitions relating to safety information see Section 10.3.

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and other safety information and remain responsible for following up AEs that are serious, considered related to study intervention or study procedures, AESIs for this study and AEs leading to discontinuation (see Section 7). This includes events reported by the participant (or, when appropriate, by a caregiver or surrogate).

The method of recording, evaluating, and assessing causality of AEs/SAEs/AESIs and the procedures for completing and transmitting SAE reports are provided in Section 10.3.

# 8.4.1. Time period and frequency for collecting AE, SAE and other safety information

All SAEs will be collected from the start of study intervention until Visit 5 at the time points specified in the SoA (Section 1.3).

SAEs assessed as related to study participation (e.g., study intervention, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product (non-IMP) will be recorded from the time a participant consents to participate in the study.

All AEs will be collected from the start of study intervention until Visit 4 at the timepoints specified in the SoA (Section 1.3).

Table 13 Timeframes for collecting and reporting of safety information

| | Screening | Dose 1 | | | | | Study Conclusion |
|---|---|---|---|---|---|---|---|
| Event | | D1 | D8 | D15 | D31 | М3 | M6 |
| Administration site and systemic solicited events* | | D 1-7 | | | | | |
| Unsolicited AEs | | | | | | | |
| | | | D1 | I-31 | | | |
| AEs/SAEs leading to withdrawal from the study | | | | | | | |
| MAAEs | | | | | | | |
| SAEs | | | | | | | |
| SAEs related to the study intervention | | | | | | | |
| SAEs related to study participation** or concurrent GSK medication/vaccine | | | | | | | |
| pIMDS | | | | | | | |
| AESIs | | | | | | | |
| Pregnancy | | | | | | | |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| | Screening | Dose 1 | | | | | Study Conclusion |
|---|---|---|---|---|---|---|---|
| Event | _ | D1 | D8 | D15 | D31 | М3 | M6 |
| Pregnancy outcomes | - | | | | | | |
| Concomitant medications | | | | | | | |

AE: Adverse events; AESI: Adverse event of special interest; D: Day, GSK: GlaxoSmithKline Biologicals SA; MAAEs: Medically attended adverse event; M: Month; pIMDs: potential Immune-mediated diseases; SAEs: Serious adverse events.

The shaded region in the table indicates time period of data collection.

<sup>\*</sup> Administration site and systemic solicited events will be collected through eDiaries.

<sup>\*\*</sup> Any SAEs assessed as related to study participation (e.g., protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product will be recorded from the time a participant consents to participate in the study.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

All SAEs will be recorded and reported to the sponsor immediately and under no circumstance should this exceed 24 hours, as indicated in Section 10.3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

A poststudy AE/SAE is defined as any event that occurs outside of the AE/SAE reporting period defined in Table 13.

Investigators are not obligated to actively seek information on AEs or SAEs after conclusion of the study participation. However, if the investigator learns of any SAE, including a death, after a participant has been discharged from the study, the investigator must record it in the medical records. If the investigator considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the sponsor.

## 8.4.2. Method of detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and SAEs. Open-ended and nonleading verbal questioning/eDiaries of the participant is the preferred method to inquire about AE occurrences.

## 8.4.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs and AESI (as defined in Section 8.4.4) will be followed until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.3). Further information on follow-up procedures is provided in Section 10.3.5.5.

#### 8.4.4. AESI

#### 8.4.4.1. pIMDs

pIMDs are a subset of AESIs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. AEs that need to be recorded and reported as pIMDs include those listed in the Table 14.

In order to facilitate the documentation of pIMDs in the eCRF, a pIMD standard questionnaire and a list of PTs and PT codes corresponding to the above diagnoses will be available to investigators at study start.

The investigator(s) must exercise their medical/scientific judgment to determine whether other diseases have an autoimmune origin (i.e., pathophysiology involving systemic or organ-specific pathogenic autoantibodies) and should also be recorded as a pIMD. In addition, the investigator should categorize each pIMD either as a new onset condition (if it started following vaccination) or as an exacerbation of a pre-existing chronic condition (if it exacerbated following vaccination) in the eCRF.

# Table 14 List of pIMDs

| Medical Concept | Additional Notes |
|---|---|
| Blood disorders and coagulopathie | |
| Antiphospholipid syndrome | |
| Autoimmune aplastic anemia | |
| Autoimmune hemolytic anemia | Includes warm antibody hemolytic anemia and cold antibody hemolytic |
| , | anemia |
| Autoimmune lymphoproliferative | |
| syndrome (ALPS) | |
| Autoimmune neutropenia | |
| Autoimmune pancytopenia | |
| Autoimmune thrombocytopenia | <ul> <li>Frequently used related terms include: "autoimmune thrombocytopenic<br/>purpura", "idiopathic thrombocytopenic purpura (ITP)", "idiopathic<br/>immune thrombocytopenia", "primary immune thrombocytopenia".</li> </ul> |
| Evans syndrome | |
| Pernicious anemia | |
| Thrombosis with | |
| thrombocytopenia syndrome (TTS) | |
| Thrombotic thrombocytopenic | Also known as "Moschcowitz-syndrome" or "microangiopathic hemolytic |
| purpura | anemia" |
| Cardio-pulmonary inflammatory dis | sorders |
| Idiopathic | Including but not limited to: |
| Myocarditis/pericarditis | Autoimmune / Immune-mediated myocarditis |
| • | Autoimmune / Immune-mediated pericarditis |
| | Giant cell myocarditis |
| Idiopathic pulmonary fibrosis | Including but not limited to: |
| , | <ul> <li>Idiopathic interstitial pneumonia (frequently used related terms include "Interstitial lung disease", "Pulmonary fibrosis", "Immune-mediated pneumonitis")</li> <li>Pleuroparenchymal fibroelastosis (PPFE)</li> </ul> |
| Pulmonary alveolar proteinosis (PAP) | Frequently used related terms include: "pulmonary alveolar lipoproteinosis", "phospholipidosis" |
| Endocrine disorders | |
| Addison's disease | |
| Autoimmune / Immune-mediated | Including but not limited to: |
| thyroiditis | <ul> <li>Hashimoto thyroiditis (autoimmune hypothyroidism, lymphocytic thyroiditis)</li> <li>Atrophic thyroiditis</li> <li>Silent thyroiditis</li> <li>Thyrotoxicosis</li> </ul> |
| Autoimmune diseases of the | Includes autoimmune oophoritis, autoimmune ovarian failure and |
| testis and ovary | autoimmune orchitis |
| Autoimmune hyperlipidemia | |
| Autoimmune hypophysitis | |
| Diabetes mellitus type I | |
| Grave's or Basedow's disease | Includes Marine Lenhart syndrome and Graves' ophthalmopathy, also known as thyroid eye disease (TED) or endocrine ophthalmopathy |
| Insulin autoimmune syndrome | |
| Polyglandular autoimmune syndrome | Includes Polyglandular autoimmune syndrome type I, II and III |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| | Protocol Amendment 3 Final |
|---|---|
| Medical Concept | Additional Notes |
| Eye disorders | |
| Ocular Autoimmune / Immune- | Including but not limited to: |
| mediated disorders | Acute macular neuroretinopathy (also known as acute macular outer |
| | retinopathy) |
| | Autoimmune / Immune-mediated retinopathy |
| | Autoimmune / Immune-mediated uveitis, including idiopathic uveitis and |
| | sympathetic ophthalmia |
| | Cogan's syndrome: an oculo-audiovestibular disease |
| | Ocular pemphigoid |
| | Ulcerative keratitis |
| | Vogt-Koyanagi-Harada disease |
| Gastrointestinal disorders | |
| Autoimmune / Immune-mediated | |
| pancreatitis | |
| Celiac disease | |
| Inflammatory Bowel disease | Including but not limited to: |
| | Crohn's disease |
| | Microscopic colitis |
| | Terminal ileitis |
| | Ulcerative colitis |
| | Ulcerative proctitis |
| Hepatobiliary disorders | |
| Autoimmune cholangitis | |
| Autoimmune hepatitis | |
| Primary biliary cirrhosis | |
| Primary sclerosing cholangitis | |
| Musculoskeletal and connective tis | |
| | Includes gouty arthritis |
| Idiopathic inflammatory | Including but not limited to: |
| myopathies | Dermatomyositis In a harism hards are saiding |
| | Inclusion body myositis |
| | Immune-mediated necrotizing myopathy Polymorphism P |
| Mind and the Air of the Air of | Polymyositis |
| Mixed connective tissue disorder | |
| Polymyalgia rheumatica (PMR) | |
| Psoriatic arthritis (PsA) | |
| Relapsing polychondritis Rheumatoid arthritis | Including but not limited to: |
| Rneumatoid artifitis | Including but not limited to: |
| | Rheumatoid arthritis associated conditions |
| | Juvenile idiopathic arthritis Palindromic rheumatism |
| | Still's disease |
| Cië avania avadana | Felty's syndrome |
| Sjögren's syndrome | Including but not limited to: |
| Spondyloarthritis | Including but not limited to: |
| | Ankylosing spondylitis Investige spondyleotheritis |
| | Juvenile spondyloarthritis Verstederme blevershading |
| | Keratoderma blenorrhagica Pagriotia anandylitia |
| | Psoriatic spondylitis Psorting Authoritie (Psitante Condenses) |
| | Reactive Arthritis (Reiter's Syndrome) Haddifferentiated and add at the fitting |
| 0.4 | Undifferentiated spondyloarthritis |
| Systemic lupus Erythematosus | Includes Lupus associated conditions (e.g., cutaneous lupus The matter of the property of the conditions of the |
| | erythematosus, lupus nephritis, etc.) or complications such as shrinking |
| | lung syndrome (SLS) |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Medical Concept | Additional Notes |
|---|---|
| Medical Concept Systemic Scleroderma (systemic | |
| sclerosis) | Includes Reynolds syndrome (RS), systemic sclerosis with diffuse Includes Reynolds syndrome (RS), systemic sclerosis with diffuse |
| scielosis) | scleroderma and systemic sclerosis with limited scleroderma (also |
| Neuroinflammatory/neuromuscular | known as CREST syndrome) |
| Acute disseminated | Includes the following: |
| encephalomyelitis (ADEM) and | |
| other inflammatory | Acute necrotizing myelitis Rickerstoff a hazinatam anaphalitis |
| demyelinating variants | Bickerstaff's brainstem encephalitis Bicagginated pagetining by languages and algorithm (alea lynguages). |
| demyemating variants | Disseminated necrotizing leukoencephalopathy (also known as Weston-Hurst syndrome, acute hemorrhagic leuko-encephalitis, or |
| | acute necrotizing hemorrhagic encephalomyelitis) |
| | Myelin oligodendrocyte glycoprotein antibody-associated disease |
| | Neuromyelitis optica (also known as Devic's disease) |
| | Noninfective encephalitis / encephalomyelitis / myelitis Partice myelitis and an encephalomyelitis |
| Cuillain Dawé aun drama (CDC) | Postimmunization encephalomyelitis |
| Guillain-Barré syndrome (GBS) | Includes variants such as Miller Fisher syndrome and the acute motor (AMOAN) (AMOAN) |
| Idionathia arenial nerve | and sensory axonal neuropathy (AMSAN) |
| Idiopathic cranial nerve | Including but not limited to: |
| palsies/paresis and inflammations (neuritis) | Cranial nerve neuritis (e.g., optic neuritis) Idiopathia para palais/passaia (e.g., Pall'a palai) |
| illiallillations (neurtus) | Idiopathic nerve palsies/paresis (e.g., Bell's palsy) Mallagrana Paragratus I and thomas |
| | Melkersson-Rosenthal syndrome Multiple special page relation/page in |
| Multiple coloresia (MS) | Multiple cranial nerve palsies/paresis |
| Multiple sclerosis (MS) | Includes the following: |
| | Clinically isolated syndrome (CIS) |
| | Malignant MS (the Marburg type of MS) By the Marburg type of MS) |
| | Primary-progressive MS (PPMS) Primary-progressive MS (PPMS) (PIG) |
| | Radiologically isolated syndrome (RIS) Reference (RIS) |
| | Relapsing-remitting MS (RRMS) |
| | Secondary-progressive MS (SPMS) |
| Musethania mavie | Uhthoff's phenomenon |
| Myasthenia gravis | Includes ocular myasthenia and Lambert-Eaton myasthenic syndrome |
| Narcolepsy | Includes narcolepsy with or without presence of unambiguous cataplexy |
| Peripheral inflammatory | Including but not limited to: |
| demyelinating neuropathies and | Acute Brachial Radiculitis (also known as Parsonage-Turner Syndrome |
| plexopathies | or neuralgic amyotrophy) |
| | Antibody-mediated demyelinating neuropathy Characteristic particles are a large property (CLAR) |
| | Chronic idiopathic axonal polyneuropathy (CIAP) Charais Inflammatica Department of Polyneuropathy (CIAP) |
| | Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP), including at visical CIDP variants (a.g., multifeed, against demyelinating). |
| | including atypical CIDP variants (e.g., multifocal acquired demyelinating sensory and motor neuropathy also known as Lewis-Sumner |
| | syndrome) |
| | Multifocal motor neuropathy (MMN) |
| Transverse myelitis (TM) | Includes acute partial transverse myelitis (APTM) and acute complete |
| Transverse myentis (Tivi) | transverse myelitis (ACTM) |
| Renal disorders | adnovoloc mychuc (no mi) |
| Autoimmune / immune-mediated | Including but not limited to: |
| glomerulonephritis | IgA nephropathy |
| <b>5</b> | IgM nephropathy |
| | C1q nephropathy |
| | Fibrillary glomerulonephritis |
| | Glomerulonephritis rapidly progressive |
| | Membranoproliferative glomerulonephritis |
| | Membranous glomerulonephritis |
| | l |
| | Tubulointerstitial nephritis and uveitis syndrome |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Madical Consent | Additional Natas |
|---|---|
| Medical Concept | Additional Notes |
| Skin and subcutaneous tissue disc | orders |
| Alopecia areata | Later Park Care Park Lie |
| Autoimmune / immune-mediated | Including but not limited to: |
| blistering dermatoses | Bullous Dermatitis |
| | Bullous Pemphigoid |
| | Dermatitis herpetiformis |
| | Epidermolysis bullosa acquisita (EBA) |
| | Linear IgA-mediated bullous dermatosis (LABD), also known as Linear |
| | lgA disease |
| | Pemphigus |
| Erythema multiforme | |
| Erythema nodosum | |
| Reactive granulomatous | Including but not limited to |
| dermatitis | Interstitial granulomatous dermatitis |
| | Palisaded neutrophilic granulomatous dermatitis |
| Lichen planus | Includes liquen planopilaris |
| Localized Scleroderma | Includes Eosinophilic fasciitis (also called Shulman syndrome) |
| (Morphoea) | |
| Psoriasis | |
| Pyoderma gangrenosum | |
| Stevens-Johnson syndrome | Including but not limited to: |
| (SJS) | Toxic Epidermal Necrolysis (TEN) |
| | SJS-TEN overlap |
| Sweet's syndrome | Includes acute febrile neutrophilic dermatosis |
| Vitiligo | |
| Vasculitis | |
| Large vessels vasculitis | Including but not limited to: |
| | Arteritic anterior ischemic optic neuropathy (AAION or arteritic AION) |
| | Giant cell arteritis (also called temporal arteritis) |
| | Takayasu's arteritis |
| Medium sized and/or small | Including but not limited to: |
| vessels vasculitis | Anti-neutrophil cytoplasmic antibody (ANCA) positive vasculitis (type |
| | unspecified) |
| | Behcet's syndrome |
| | Buerger's disease (thromboangiitis obliterans) |
| | Churg–Strauss syndrome (allergic granulomatous angiitis) |
| | Erythema induratum (also known as nodular vasculitis) |
| | Henoch-Schonlein purpura (also known as IgA vasculitis) |
| | Microscopic polyangiitis |
| | Necrotizing vasculitis |
| | Polyarteritis nodosa |
| | Single organ cutaneous vasculitis, including leukocytoclastic vasculitis, |
| | hypersensitivity vasculitis and acute hemorrhagic edema of infancy |
| | (AHEI) |
| | Wegener's granulomatosis |
| Other (including multisystemic) | |
| Anti-synthetase syndrome | |
| Capillary leak syndrome | Frequently used related terms include "systemic capillary leak (2010)" "(2011)" "(2011) |
| 01 | syndrome (SCLS)" or "Clarkson's Syndrome" |
| Goodpasture syndrome | Frequently used related terms include "pulmonary renal syndrome" and |
| - Cocapactaro cyrrar crist | "anti-Glomerular Basement Membrane disease (anti-GBM disease)" |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Medical Concept | Additional Notes |
|---|---|
| Immune-mediated enhancement of disease | <ul> <li>Includes vaccine associated enhanced disease (VAED and VAERD). Frequently used related terms include "vaccine-mediated enhanced disease (VMED)", "enhanced respiratory disease (ERD)", "vaccine-induced enhancement of infection", "disease enhancement", "immune enhancement", and "antibody-dependent enhancement (ADE) </li> </ul> |
| Immunoglobulin G4 related disease | |
| Langerhans cell histiocytosis | |
| Multisystem inflammatory syndromes | Including but not limited to: <ul> <li>Kawasaki's disease</li> <li>Multisystem inflammatory syndrome in adults (MIS-A)</li> <li>Multisystem inflammatory syndrome in children (MIS-C)</li> </ul> |
| Overlap syndrome | |
| Raynaud's phenomenon | |
| Sarcoidosis | Includes Loefgren syndrome |
| Susac's syndrome | |

IgA: Immunoglobulin A; IgM: Immunoglobulin M.

#### 8.4.4.2. Other AESIs

- Myocarditis and pericarditis
- Virologically confirmed COVID-19 cases
- Anaphylaxis or severe hypersensitivity within 24 hours after study vaccination

When there is enough evidence to make any of the above diagnoses, the AE must be reported as AESI. Symptoms, signs or conditions which might (or might not) lead to one of the above diagnoses, should be recorded and reported as AEs but not as AESI until the final or definitive diagnosis has been made, and alternative diagnoses eliminated or shown to be less likely.

#### 8.4.4.2.1. Myocarditis and pericarditis: definitions and assessment

All potential cases of myocarditis and pericarditis will be provided to the independent external adjudication committee for case adjudication according to the case definition from the Brighton Collaboration [Sexson, 2022].

Source documentation of suspected cases of myocarditis and pericarditis to be provided for adjudication as it becomes available may include (but are not limited to) the following:

- Clinical notes (including history, physical examination, EKG findings)
- Emergency department notes (including history, physical examination, EKG findings)
- Hospital discharge summary
- Clinical laboratory values
- Concomitant medications

- Chest X-ray reports
- Cardiac imaging

Following adjudication, all probable and definitive cases of myocarditis and pericarditis will be reviewed by SRT (blinded data review until Part A Day 15 interim analysis, unblinded data review subsequently) and iSRC (unblinded data review). An ad-hoc iSRC will be conducted on receiving any probable or definitive cases of myocarditis and pericarditis. An independent external cardiologist may be part of iSRC to provide input on the potential myocarditis and pericarditis cases.

### Clinical myocarditis/pericarditis:

The participants reporting acute chest pain, shortness of breath or other signs/symptoms of myocarditis/pericarditis within 6 weeks after vaccination must be evaluated by a cardiologist with evaluation and management following current practice guidelines (e.g., American heart association or local standard of care).

The changes suggestive of myocarditis and pericarditis (but not limited to) are listed below:

- EKG changes:
  - ST segment or T wave abnormalities (elevation or inversion)
  - Paroxysmal or sustained atrial or ventricular arrhythmias
  - AV nodal conduction delays or intraventricular conduction defects.
  - An abnormal troponin I value (> 2 ULN of baseline value) that is confirmed abnormal on repeat testing.
- Cardiac imaging:
  - Echocardiogram: New left or right ventricular function abnormalities including: segmental wall motion abnormalities; decreased ejection fraction (EF <55% for ≤54 yrs; or <50% for >55 yrs); global systolic or diastolic function depression/abnormality; ventricular dilation or wall thickness change; pericardial effusion or intracavitary thrombi
  - Cardiac MRI: Patchy edema on T2 weighted images or late gadolinium enhancement on T1 weighted images with increased enhancement ratio between myocardial skeletal muscle involving ≥1 non-ischemic regional distribution with recovery

The participants will be followed-up until the resolution of symptoms and/or cardiac troponin levels return back to normal.

#### Asymptomatic myocarditis/pericarditis:

At the Day 8 (Visit 2), all participants will be assessed by 12-lead EKG for evidence of asymptomatic myocarditis or pericarditis, based on evidence that rare cases of myocarditis or pericarditis have occurred most frequently within 7 days of vaccination
219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

[CDC, 2023]. All participants will also have a 12-lead EKG examination at screening, to provide a baseline for comparison.

Asymptomatic acute myocarditis/pericarditis is defined as electrocardiographic changes suggestive of acute myocardial injury occurring in an asymptomatic participant within 6 weeks after administration of a COVID-19 mRNA vaccine, if other causes of acute cardiac disease are excluded. If any of the EKG changes suggestive of myocarditis and pericarditis listed above are detected at the surveillance EKG occurring at the Day 8 visit, the findings will be reviewed by the investigator.

If deemed appropriate the participant will be referred to a local cardiologist. If a diagnosis of myocarditis or pericarditis is confirmed, then the participant will be further evaluated and receive cardiology consultation, including cardiac enzyme assessment, echocardiography, or other assessments deemed clinically warranted by the treating clinician.

## 8.4.4.2.2. SARS-CoV-2 infection and COVID-19 definitions and assessment

Vaccine efficacy will not be evaluated in this study, but all laboratory-confirmed asymptomatic SARS-CoV-2 infections should be reported by the participant and documented as AEs, while virologically confirmed cases of COVID-19 are reported as AESIs. Any available isolate genotyping results will also be requested. Participants will be instructed to inform the investigator in the event of a positive SARS-CoV-2 diagnostic test. Serology testing for SARS-CoV-2 N protein will be performed pre-vaccination and post-vaccination to monitor for undetected SARS-CoV-2 infections at the time points specified in the SoA (Section 1.3).

All participants with suspected COVID-19 are required to have an unscheduled visit for suspected COVID-19, as detailed in the SoA (Section 1.3). At this visit, participants will undergo the following assessments:

- Medical history
- SARS-CoV-2 RT-PCR (nasopharyngeal or mid-turbinate swab)
- Physical examination
- Vital sign measurements
- Body temperature
- Review of AEs
- Concomitant medication/vaccination

All participants with confirmed COVID-19 are required to have an unscheduled COVID-19 convalescent visit as detailed in the SoA (Section 1.3). At this visit, participants will undergo the following assessments:

- Medical history
- SARS-CoV-2 RT-PCR (nasopharyngeal or mid-turbinate swab)

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- Physical examination
- Vital sign measurements
- Body temperature
- COVID-19 evaluation
- Review of AEs
- Concomitant medication/vaccination

To complete the COVID-19 evaluation, the investigator will review the history of the participants, including medical records to define the severity of COVID-19.

Any confirmed cases of SARS-CoV-2 infection or COVID-19 during the study will be assigned one of the following definitions and recorded in the eCRF:

Asymptomatic SARS-CoV-2 infection:

Laboratory-confirmed SARS-CoV-2 by RT-PCR or SARS-CoV-2 N protein seroconversion without any of the following symptoms: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea

COVID-19:

Virologically confirmed SARS-CoV-2 by RT-PCR with 1 or more of the following symptoms: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea

Severe COVID-19:

Virologically confirmed SARS-CoV-2 infection with any 1 of the following:

- Clinical signs at rest indicative of severe systemic illness (respiratory rate ≥ 30 per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300 mm Hg)
- Respiratory failure (defined as needing high-flow oxygen, non-invasive ventilation, mechanical ventilation, or ECMO)
- Evidence of shock (systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg, or requiring vasopressors)
- Significant acute renal, hepatic, or neurologic dysfunction
- Admission to a hospital or an intensive care unit
- Death

## 8.4.5. Regulatory reporting requirements for SAEs/AESIs

- Prompt notification by the investigator to the sponsor of an SAE/AESI is essential so
  that legal obligations and ethical responsibilities toward the safety of participants and
  the safety of a study intervention under clinical investigation are met. See
  Section 8.4.1 for reporting timeframes.
- For SAEs/AESIs, the investigator must always provide an assessment of causality at the time of the initial report, as defined in the Section 10.3.5.3.
- An investigator who receives an investigator safety report describing an SAE or other specific safety information (e.g., summary or listing of SAEs) from the sponsor will review and then file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.
- Once an investigator (or designee) becomes aware that a study participant has
  experienced an SAE/AESI/pregnancy, it must be reported to the CRO medical
  monitor using the required documentation and within the timeframes mentioned in
  Table 15. This is essential for GSK to meet legal obligations and ethical
  responsibilities for participant safety and the safety of a study intervention under
  clinical investigation.
- The sponsor has the legal responsibility to notify local authorities/regulatory agencies about the safety of an investigational study intervention. The sponsor will comply with country-specific regulatory requirements related to safety reporting to the regulatory authority, IRB/IEC and investigators.
- Please refer to Section 10.3.5.7 for further details regarding the reporting of SAEs/AESIs/pregnancies.

Table 15 Timeframes for submitting SAE, AESI, pregnancy and other events reports to CRO

| Type of event | Initial reports | | Follow-up of relevant information on a previous report | |
|---|---|---|---|---|
| | Timeframe | Documents | Timeframe | Documents |
| SAEs | 24 hours* ## electronic AE report | | 24 hours* | electronic AE report |
| Pregnancies | 24 hours* electronic pregnancy report | | 24 hours * | electronic pregnancy report |
| AESIs | 24 hours** ‡‡ electronic AE report | | 24 hours* | electronic AE report |

AE: Adverse event; Adverse event of special interest; SAE: Serious adverse event.

## 8.4.6. Pregnancy

Female participants who become pregnant after administration of the study intervention may continue the study at the discretion of the investigator.

• Details of all pregnancies in female participants will be collected after the start of study intervention and until Day 31.

<sup>\*</sup> Timeframe allowed after receipt or awareness of the information by the investigator/site staff.

<sup>\*\*</sup>Timeframe allowed once the investigator determines that the event meets the protocol definition of an AESI.

<sup>&</sup>lt;sup>‡‡</sup> For each SAE/AESI, the investigator(s) must document in the medical notes that they have reviewed the SAE/AESI and have provided an assessment of causality.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- If a pregnancy is reported, the investigator will record pregnancy information on the appropriate form and submit it to the sponsor within 24 hours of learning of the female participant pregnancy.
- Any pregnancy complication or elective termination of a pregnancy for medical reasons will be reported as an AE or SAE.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs and will be reported as such.
- The participant will be followed to determine the outcome of the pregnancy. The investigator will collect follow-up information on the participant/pregnant female partner and the neonate and the information will be forwarded to the sponsor. See Table 15 for reporting timeframes.
- Any poststudy pregnancy-related SAE considered reasonably related to the study intervention by the investigator will be reported to the sponsor as described in Section 10.3.5.7. While the investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.

# 8.4.7. Contact information for reporting SAEs, AESIs, pregnancies and study holding rules

Table 16 Contact information for reporting SAEs, AESIs, pregnancies and study holding rules

| Study contact for questions regarding SAEs, AESIs, pregnancies | Study contact for reporting of study holding rules |
|---|---|
| If a SAEs, AESIs, pregnancies are reported, the investigator must inform the CRO medical monitor | If a holding rule is met, the investigator must immediately inform the CRO medical monitor. |
| Back up study contact for reporting SAEs, AESIs, pregnancies | Back up study contact for escalation of holding rules |
| Available 24/24 hours and 7/7 days: | Available 24/24 hours and 7/7 days: |
| CRO hotline | |
| North America: | |
| +1 800 201 8725 (phone) | |
| +1 888 488 9697 (fax) | |

76

## 8.4.8. Participant card

The investigator (or designee) must provide the participant with a "participant card" containing information about the clinical study. The participant must be instructed to always keep the participant card in their possession for the duration of the study. In an emergency, this card serves to inform the responsible attending physician that the participant is in a clinical study and that relevant information may be obtained by contacting the investigator(s).

## 8.5. Pharmacokinetics

Not applicable.

## 8.6. Genetics

Not applicable.

## 8.7. Biomarkers

Not applicable.

## 8.8. Immunogenicity assessments

Immunogenicity is described in Section 8.2.

## 8.9. Health outcomes

Not applicable.

## 8.10. Study procedures during special circumstances

During special circumstances (e.g., COVID-19 pandemic), the specific guidance from local public health and other competent authorities regarding the protection of individuals' welfare must be applied. For the duration of such special circumstances, the following measures may be implemented for enrolled participants:

- Further in-person clinic visits may be suspended.
- Safety follow-up may be made by a telephone call, other means of virtual contact or home visit, if appropriate.
- If the eDiary device was provided to the participant, it may be returned to the site by conventional mail after the end of the safety period for collection of solicited events following Visit 2 (Day 8), inclusive of the allowable window period).

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- Visits for suspected COVID-19 may take place in a different location\* other than the study site or at participant's home. If this is not feasible, then the medical evaluation of COVID-19 may take place virtually with documentation of event by telephone/telemedicine.
- Biological samples may be collected at a different location\* other than the study site or at participant's home. Biological samples should not be collected if they cannot be processed in a timely manner or appropriately stored until the intended use.

\*It is the investigator's responsibility to identify an alternate location. The investigator should ensure that this alternate location meets ICH GCP requirements, such as adequate facilities to perform study procedures, appropriate training of the staff and documented delegation of responsibilities in this location. This alternate location should be covered by proper insurance for the conduct of study on participants by investigator and staff at a site other than the designated study site. Refer to the EMA guidance on the management of clinical trials during the COVID-19 (Coronavirus) pandemic (version 2, 27 March, 2020) for more details.

Impact on the PPS for immunogenicity will be determined on a case-by-case basis.

## 9. STATISTICAL CONSIDERATIONS

## 9.1. Statistical hypotheses

There is no hypothesis testing in this study; all analysis will be performed in a descriptive manner. Means and proportions for different objectives will be computed with their 95% CIs.

## 9.2. Sample size determination

The sample size is based on clinical considerations to inform dose regimen decisions for continued clinical development.

With 18 participants receiving mRNA-CR-04 vaccine in each group, there is a 60.3% probability to observe at least 1 AE if the incidence rate is 5% and 85% probability to observe at least 1 AE if the incidence rate is 10%.

With 16 participants receiving mRNA-CR-04 vaccine in each group (PPS for immunogenicity, 10% unevaluable), and a standard deviation of 0.45 for log<sub>10</sub> transformed increase from Day 1, the ratio of the upper limit of a 2-sided 95% CI and the point estimate of GMR is 1.74.

## 9.3. Analysis sets

Table 17 Analysis sets

| Analysis set | Description |
|---|---|
| Screened | All participants who were screened for eligibility. |
| Enrolled | Participants who completed the informed consent process, meet screening/eligibility criteria and undergone an invasive procedure. Note: screening failures (who never passed screening even if re-screened) and participants screened but never enrolled into the study (Met eligibility but not needed) are excluded from the Enrolled analysis set as they did not enter the study. |
| Exposed | All participants who received the dose of the study intervention. Analysis per group using the enrolled set based on the administered intervention. |
| Per Protocol | All eligible participants who received dose of study intervention as per protocol, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination, and who have values for pre-dose and post-dose neutralizing antibody titer against pseudovirus bearing S protein data for the relevant timepoint, and without major protocol deviations. The PPS for immunogenicity will be defined by time point. |
| Solicited Safety | All participants who received the dose of the study intervention (Exposed Set) who have reported the presence or absence of any solicited AE at least once. |

AE: Adverse event; D: Day; S: Spike; PPS: Per Protocol Set

## 9.3.1. Criteria for elimination from analysis

If a participant meets one of the criteria mentioned below, they may be eliminated from per protocol analysis.

- Receive any of the medications/products/vaccines listed in Section 5.2.2.
- Incur an intercurrent medical condition that could alter their immune response (i.e., varicella, HIV, lymphoma) or are confirmed to have an alteration of their initial immune status.
- Major protocol deviation(s) linked to the eligibility criteria (Section 5.1 and Section 5.2).
- Study intervention not administered as specified by the protocol.
- Failure to comply with the post-dose immunogenicity blood sampling schedule at a given timepoint (Section 1.3).
- Other major protocol deviation during vaccination phase that led to exclusion.

The SAP will provide a complete list of criteria for elimination from PP analyses.

## 9.4. Statistical analyses

The SAP will be finalized prior to FSFV and it will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints including primary and secondary endpoints.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

For the vendors that will perform statistical activities, please refer to the separate list of vendors for details.

## 9.4.1. Primary endpoint

Analysis of primary safety endpoints will be performed on the Exposed Set, except for solicited AEs, which will be performed on the Solicited Safety Set. The analysis will be performed separately for study Part A and Part B participants. In addition, pooled analyses where groups common in Part A and Part B are combined as one group respectively will be performed.

## Statistical analysis methods

The number and percentage of participants reporting AEs up to 30 days after the dose (Day 31):

- At least one administration site event (solicited and unsolicited), with at least one systemic event (solicited and unsolicited) and with any AE (solicited and unsolicited) during the 7-day and 30-day follow-up period will be tabulated by treatment. Same tabulations will be performed for Grade 3 AEs (all and causally related) and for any causally related AEs.
- Each individual solicited administration site event (any grade and Grade 3) and solicited systemic event (any grade and Grade 3) during the 7-day follow-up period will be tabulated by maximum intensity per participant for each treatment group.
- Fever will be reported as number and percentage of participants reporting temperature per 0.5°C cumulative increments as from ≥38°C or 100.4°F during the 7-day follow-up period (i.e., on the day of study intervention administration and 6 subsequent days) and will be tabulated for each treatment group.
- At least one unsolicited AE during the 30-day follow-up period after the dose, as classified by the MedDRA SOC and PT will be tabulated by treatment group. The same tabulation will be performed for Grade 3, any causally related, Grade 3 causally related unsolicited AEs and unsolicited AEs with medically attended visits.
- For each treatment group and for each hematology and biochemistry parameter:
  - The number and percentage of participants having hematology and biochemistry results below or above the laboratory normal ranges will be tabulated by time point.
  - The maximum grading post-dose up to Day 15 will be tabulated versus baseline (Day 1, or if not available, closest visit available to D1 before IMP administration). Grades will be based on the FDA guidance for industry "Toxicity grading scale for healthy adults and adolescent volunteers enrolled in preventive vaccine clinical trials" (Section 10.2.2).
- At least one MAAE, SAE and AESIs after the dose, as classified by the MedDRA SOC and PT, will be tabulated by treatment group. The same tabulation will be performed for causally related MAAEs, SAEs and AESIs during this period. The detailed listings of SAEs, AESIs and COVID-19 cases will also be produced.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

• At least one concomitant medication (any medication or any antipyretic) during the 7-day follow-up period and during the 30-day follow-up will be summarized by treatment group.

## 9.4.2. Secondary endpoints/estimands analyses

## 9.4.2.1. Safety endpoints

Analysis of secondary safety endpoints will be performed on the Exposed Set. The analysis will be performed separately for study Part A and Part B participants. In addition, pooled analyses where groups common in Part A and Part B are combined as one group respectively will be performed.

## Statistical analysis methods

The number and percentage of participants with AEs up to study conclusion (Month 6):

- At least one MAAE, SAE and AESIs after the dose, as classified by the MedDRA SOC and PT, will be tabulated by treatment group. The same tabulation will be performed for causally related MAAEs, SAEs and AESIs during this period. The detailed listings of SAEs, AESIs and COVID-19 cases will also be produced.
- A listing of AEs/SAEs leading to withdrawal from the study will be provided.

## 9.4.2.2. Immunogenicity endpoints

The analysis of the secondary immunogenicity endpoints will be performed on the PPS separately for study Part A and Part B participants. In addition, pooled analyses where groups common in Part A and Part B are combined as one group respectively will be performed. If more than 10% of participants are eliminated from any of the PPS in any treatment group, a sensitivity analysis will be carried out using the Exposed Set.

## Statistical analysis methods

Following **humoral immune responses** (neutralizing titer) will be summarized by treatment group using descriptive statistics, using corresponding blood sample collected for assessment of humoral immune responses:

- Neutralizing titer (GMT) against pseudovirus bearing S protein from vaccine encoded SARS-CoV-2 and WT strains will be tabulated with 95% CI and represented graphically.
- GMR from baseline of neutralizing titer against pseudovirus bearing S protein from vaccine encoded SARS-CoV-2 and WT strains at each collection time point after administration of study intervention over time point before administration of study intervention will be tabulated with 95% CI.
- GMTs and GMRs from baseline of neutralizing titer, with their 95% CI, using an ANCOVA on log-transformed titer with treatment group as a fixed factor, and Day 1

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

baseline value as a covariable. GMTs and GMRs will also be represented graphically. Once Part B data are available, Part A and Part B data will be pooled together for model based analyses. When pooled, the study part will be added as a fixed factor and adjusted GMT/GMR will be estimated under Part A condition. Groups common in Part A and Part B will be combined as one group respectively for the pooled analysis.

• Percentage of participants with vaccine responses of a 4-fold increase from Day 1, with their exact 95% CI will be tabulated.

## 9.4.3. Analyses of exploratory immunogenicity endpoints

Additional exploratory immunological assays evaluating S-specific or disease-related antigen specific humoral or cellular immune responses, including but not limited to antibody functionality (Fc $\gamma$  R binding capacity, IgG affinity), isotype titer and isotype avidity, deep immunophenotyping of cellular responses might also be performed. The analyses will be performed separately for study Part A and Part B participants. In addition, pooled analyses where groups common in Part A and Part B are combined as one group respectively will be performed. Appropriate pooled analyses, such as the ANCOVA planned on neutralizing antibody titers will also be performed on the IgG antibody responses.

Analysis of tertiary endpoints detailed in Section 3 will be described in the SAP.

## 9.5. Interim analyses

No interim analysis requiring statistical adjustment will be performed. However, analyses to evaluate objectives and endpoints will be performed in steps. The sequence of analyses is described below.

## 9.5.1. Sequence of analyses

- In preparation of the safety review during the dose-escalation safety lead-in, analyses of available safety data will be performed
- Day 15 interim analysis for each group in Part A of the study will include all the data (Day 1 and Day 15) pertaining to primary and secondary safety; humoral immunogenicity (including at least neutralizing titer against pseudovirus bearing S protein from vaccine encoded SARS-COV-2 endpoints). This analysis will be performed when all data of each study group up to Day 15 (i.e., data that are as clean as possible) are available.
  - Results of this analysis will be presented in a Day 15 statistical analysis report.
  - This analysis will be performed by independent unblinded statistician who will be unblinded for this analysis, who will generate a statistical report by treatment group but no individual listings.
    - The investigators and study participants will stay blinded (i.e., will not have access to the individual participant treatment assignment) until EoS.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- A similar to Part A Day 15 interim analysis for participants in Part B of the study may be conducted separately or incorporated into a Day 31 interim analysis.
- Day 31 interim analysis for each group in Part A of the study will include all the data (Day 1, Day 15, and Day 31) pertaining to primary and secondary safety; humoral immunogenicity (including at least neutralizing titer against pseudovirus bearing S protein from vaccine encoded SARS-COV-2 endpoints). This analysis will be performed when all data of each study group up to Day 31 (i.e., data that are as clean as possible) are available.
  - Results of this analysis will be presented in a Day 31 statistical analysis report.
  - The investigators and study participants will stay blinded (i.e., will not have access to the individual participant treatment assignment) until EoS.
- A similar to Part A Day 31 interim analysis for participants in Part B of the study may be conducted separately or incorporated into the final analysis.
- The final analysis will include all the data pertaining to primary and secondary safety and immunogenicity endpoints, and any available tertiary endpoint(s). This analysis will be performed at the EoS when all data up to study conclusion (Month 6) are available. This includes Day 1, Day 15, Day 31, and Month 6, as all the data analyzed in the Day 15 and Day 31 analyses will be included in the final analysis as well.

The final study report will contain at least the final analyses of all primary and secondary endpoints, including individual listings.

If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These analyses will be documented in annex(es) to the study report.

## 9.5.2. Statistical consideration for Interim analyses

Not applicable.

# 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

## 10.1. Appendix 1: Regulatory, ethical, and study oversight considerations

## 10.1.1. Regulatory and ethical considerations

- This study will be conducted in accordance with the protocol and with:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and CIOMS International Ethical Guidelines
  - Applicable ICH GCP Guidelines

- Applicable laws and regulations
- The protocol, protocol amendments, ICF, IB, and other relevant documents (e.g., eDiary) must be submitted to an IRB/IEC by the investigator for review and approval. These documents will be signed and dated by the investigator before the study is initiated.
- Any protocol amendments will require IEC/IRB approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- GSK will provide full details of the above procedures to the investigator, either verbally, in writing, or both.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually
    or more frequently in accordance with the requirements, policies, and
    procedures established by the IRB/EC.
  - Notifying the IRB/IEC of SAE(s) or other significant safety findings as required by IRB/IEC procedures.
  - Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations.

## 10.1.2. Financial disclosure

Investigators and sub-investigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the study and for 1 year after completion of the study.

## 10.1.3. Informed consent process

The investigator(s) or their representative(s) must fully explain the nature of the study to the participant and answer all questions regarding the study.

Participants must be informed that their participation is voluntary.

Freely given and written informed consent must be obtained from each participant, as appropriate, prior to participation in the study.

The content of the ICF must meet the requirements of 21 CFR 50, local regulations, ICH guidelines, HIPAA requirements, privacy and data protection requirements, where applicable, and the IRB/IEC or study center.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.

Participants must be re-consented to the most current version of the ICF(s) or an ICF addendum during their participation in the study.

In case of unexpected pregnancy, participant must be informed that PI such as the date of birth and sex of the baby will be collected as part of safety follow-up. Consent for the baby may be obtained from the participant and/or their partner as per local regulations.

A physical or digital copy of the ICF must be provided to the participants.

Participants who are re-screened are required to sign a new ICF.

## 10.1.4. Data protection

Participants will be assigned a unique identifier by the investigator. Any participant records or datasets transferred to the sponsor will contain only the identifier. Name and any other information which would identify the participant will not be transferred.

GSK will ensure protection of the personal data of the investigator and site staff which is collected within the framework of and for the purpose of the study.

The participants must be informed that:

- Their personal study-related data will be used by the sponsor in accordance with local data protection law.
- Their medical records may be examined by clinical quality assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

The participants must be notified about their rights regarding the use of their personal data in accordance with the data privacy section of the ICF.

## 10.1.5. Committees structure

The study will be overseen by an SRT, and iSRC operating under a charter.

The SRT is an internal team, with representatives of different functions (including safety physician, a CSL and a biostatistician) involved in the conduct of the study/project.

A SRT is in place for each GSK product. It comprises of a global cross-functional team responsible for the ongoing assessment of benefit-risk for a product. The SRT contribute to the continual assessment of incoming new efficacy and safety information.

The iSRC is an internal committee including a GSK safety physician, a CSL and a biostatistician who are not otherwise involved in the conduct of the project.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

More details on the composition, objectives, and responsibilities of the iSRC will be described in the charter.

Furthermore, to enhance independent, systematic, and standardized identification, processing and review of probable or confirmed cases of myocarditis or pericarditis; an independent external cardiologist will review and assess all performed EKGs (Screening, Day 8, unscheduled visits) and an independent adjudication committee will perform case adjudication according to the case definition from the Brighton Collaboration [Sexson, 2022]. Details of data collection and frequency of data review are provided in Section 8.4.4.2.1.

## 10.1.6. Dissemination of clinical study data

The key design elements of this protocol and results summaries will be posted on www.ClinicalTrials.gov and/or GSK clinical study register in compliance with applicable regulations/GSK policy. GSK will aim to register protocols summaries prior to study start and target results summaries submission within 12 months of primary/study completion date. Where external regulations require earlier disclosure, GSK will follow those timelines.

Where required by regulation, summaries will also be posted on applicable national or regional clinical study registers.

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the study report, and provided reasonable access to statistical tables, figures, and relevant reports. GSK will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study participants, as appropriate.

GSK will provide the investigator with the randomization codes for their site only after completion of the full statistical analysis.

GSK intends to make anonymized patient-level data from this study available to external researchers for scientific analyses or to conduct further research that can help advance medical science or improve patient care. This helps ensure the data provided by study participants are used to maximum effect in the creation of knowledge and understanding.

## 10.1.7. Data quality assurance

The investigator should maintain a record of the location(s) of their respective essential documents, including source documents (see Definition of terms for the exact definition of essential and source documents). The document storage system used during the study and for archiving (irrespective of the type of media used) should provide for document identification, version history, search, and retrieval.

Essential study documents may be added or removed where justified (in advance of study initiation) based on their importance and relevance to the study. When a copy is used to replace an original document (e.g., source documents, CRF), the copy should fulfill the

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

requirements for certified copies (see Definition of terms for the exact definition of certified copies).

All participant data related to the study will be recorded on printed or electronic CRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF.

The investigator must maintain adequate and accurate source documents and study records that include all pertinent observations on each of the site's study participants (see Definition of terms for the exact definition of source documents) that supports information entered in the eCRF.

The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source documents or certified copies for such review and inspection.

The sponsor or designee is responsible for the data management of this study including quality checking of the source data (see Definition of terms for the exact definition of source data).

Study monitors will perform ongoing source data verification to confirm that data entered in the eCRF by authorized site personnel are attributable, legible, contemporaneous, original, accurate, and complete. Changes to source data must be traceable, not obscure the original entry, and be fully explained if necessary (e.g., via an audit trail). The safety and rights of participants must be protected, and the study conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

QTLs will be pre-defined in the centralized monitoring plan to identify systematic issues that can impact participant safety and/or the reliability of study results. These pre-defined parameters will be monitored during the study. Important deviations from the QTLs and remedial actions taken will be summarized in the CSR.

Study records and source documents pertaining to the conduct of this study, including signed ICFs, must be retained by the investigator for 25 years from issuance of the final CSR/equivalent summary unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

When copies of source documents are shared externally for review by a central reader mechanism (e.g., independent external cardiologist, adjudication committee), documents are stored by the external body for approximately 3 years.

## 10.1.8. Source documents

Source documents provide evidence to establish the existence of the participant and substantiate the integrity of collected data. The investigator should maintain a record of the location(s) of their source documents.

Data transcribed into the eCRF from source documents must be consistent with those source documents; any discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

Definitions of what constitutes source data and documents can be found in the Definition of terms.

Copies of documents are shared with external third parties contracted by GSK for review by a central reader mechanism (e.g., independent external cardiologist, adjudication committee). The non-exhaustive list of documents shared to inform the central reader may include EKG reports, lab data, medical records etc. Participant names or any information which would make the participant identifiable or is not essential for the central reader mechanism will be redacted prior to transfer. Details of the list of documents and the redaction procedure are provided in the site manual or equivalent. These documents will be used by the third party solely for the purpose indicated within this protocol.

## 10.1.9. Study and site start and closure

#### First act of recruitment

The start of study is defined as FSFV at a country-level.

## Study/Site termination

GSK or its designee reserves the right to close the study site or terminate the study at any time for any reason at its sole discretion, provided there is sufficient notice given to account for all participants safe exit from study.

Regular closure of study sites will occur upon study completion. A study site is considered closed when all required data/documents and study supplies have been collected and a study site closure visit has been performed.

The investigator may initiate study site closure at any time, provided there is reasonable cause and enough notice in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

• Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines

- Inadequate recruitment of participants by the investigator
- Discontinuation of further study intervention development
- Total number of participants included earlier than expected

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the IECs/IRBs, the regulatory authorities, and any CRO(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

## 10.1.10. Publication policy

GSK aims to submit the results of the study for publication in searchable, peer reviewed scientific literature within 18 months from the LSLV for interventional studies and follows the guidance from the ICMJE.

## 10.2. Appendix 2: Clinical laboratory tests

## 10.2.1. Protocol required safety laboratory assessments

The tests detailed in Table 18 will be performed by the CRO PPD.

Table 18 Protocol required safety laboratory assessments

| Laboratory assessments | Parameters | | | |
|---|---|---|---|---|
| Hematology | Platelet Count RBC Count Hemoglobin Prothrombin Time / INR | RBC Indices: MCV MCH %Reticulocytes | | WBC count with differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils |
| Clinical chemistry | BUN | | AST | Total and direct bilirubin |
| | Creatinine | | ALT | |
| | | | ALP | |
| Other tests | Follicle stimulating hormone (as needed in WONCBP only) Cardiac troponin (troponin I) [Serum or urine hCG pregnancy test (as needed for WOCBP)] The results of each test carried out locally must be entered in the eCRF. | | | |

#### NOTES:

All events of ALT  $\ge 3x$  ULN AND total bilirubin  $\ge 2x$  ULN (>35% direct bilirubin) or INR >1.5, which may indicate severe liver injury (possible Hy's Law), must be reported as an SAE.

All events of Troponin  $I \ge 2$  x baseline value, may require clinical review.

Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.

ALP: Alkaline phosphatase; ALT: Alanine aminotransferase; AST: Aspartate aminotransferase; BUN: Blood urea nitrogen; eCRF: electronic Case report form; hCG: human Chorionic gonadotropin; INR: International normalized ratio; IEC: Independent ethics committee; IRB: Institutional review board; MCH: Mean corpuscular hemoglobin; MCV: Mean corpuscular volume; RBC: Red blood cell; SAE: Serious adverse event; ULN: upper limit of normal; WBC: White blood cell; WONCBP: Woman of non-child-bearing potential; WOCBP: Woman of childbearing potential.

89

# 10.2.2. Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials

The laboratory values provided in the tables below serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

Table 19 Toxicity grading scales for biochemistry parameters evaluated in the current study\*

| Serum ** | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) | Potentially life<br>threatening<br>(Grade 4)*** |
|---|---|---|---|---|
| BUN mg/dL | 23 – 26 | 27 – 31 | > 31 | Requires dialysis |
| Creatinine mg/dL | 1.5 – 1.7 | 1.8 – 2.0 | 2.1 – 2.5 | > 2.5 or requires dialysis |
| Liver function tests –<br>ALT, AST<br>increase by factor | 1.1 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| ALP – increase by factor | 1.1 – 2.0 x ULN | 2.1 – 3.0 x ULN | 3.1 – 10 x ULN | > 10 x ULN |
| Bilirubin – when liver function test is normal; increase by factor | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| Bilirubin – when accompanied by any increase in liver function test increase by factor | 1.1 – 1.25 x ULN | 1.26 – 1.5 x ULN | 1.51 – 1.75 x ULN | > 1.75 x ULN |

ALP: Alkaline phosphatase; ALT: Alanine aminotransferase; AST: Aspartate aminotransferase; BUN: Blood urea nitrogen; ULN: upper limit of normal.

<sup>\*</sup> Toxicity grading taken from FDA guidance for industry: Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials [FDA, 2007].

<sup>\*\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

<sup>\*\*\*</sup> The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as potentially life-threatening (Grade 4). For example, a low sodium value that falls within a Grade 3 parameter (125-129 mE/L) should be recorded as a Grade 4 hyponatremia event if the participant had a new seizure associated with the low sodium value.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Table 20 Toxicity grading scales for hematology parameters evaluated in the current study\*

| Hematology** | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially life-<br>threatening<br>(Grade 4) |
|---|---|---|---|---|
| Hemoglobin (Female) - gm/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | < 8.0 |
| Hemoglobin (Female)<br>change from baseline<br>value - gm/dL | Any decrease –<br>1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| Hemoglobin (Male) - gm/dL | 12.5 – 13.5 | 10.5 – 12.4 | 8.5 – 10.4 | < 8.5 |
| Hemoglobin (Male)<br>change from baseline<br>value – gm/dL | Any decrease –<br>1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| WBC Increase - cell/mm <sup>3</sup> | 10,800 – 15,000 | 15,001 – 20,000 | 20,001 – 25,000 | > 25,000 |
| WBC Decrease - cell/mm <sup>3</sup> | 2,500 – 3,500 | 1,500 – 2,499 | 1,000 – 1,499 | < 1,000 |
| Lymphocytes decrease - cell/mm <sup>3</sup> | 750 – 1 000 | 500 – 749 | 250 – 499 | < 250 |
| Neutrophils decrease - cell/mm <sup>3</sup> | 1,500 – 2,000 | 1,000 – 1,499 | 500 – 999 | < 500 |
| Eosinophils - cell/mm <sup>3</sup> | 650 – 1 500 | 1,501 – 5,000 | > 5,000 | Hypereosinophilic |
| Platelets decreased - cell/mm <sup>3</sup> | 125,000 – 140,000 | 100,000 – 124,000 | 25,000 – 99,000 | < 25,000 |
| Prothrombin Time – increase by factor | 1.03 – 1.10 x ULN | 1.11 – 1.20 x ULN | 1.21 – 1.25 x ULN | >1.25 x ULN |

ULN: Upper limit of the normal range; WBC: White blood cell.

In order to determine the grading, the following rules will be used:

- 1. In case a conversion is needed, the original results will be used for the conversion without a previous rounding.
- 2. In case an approximation is needed to determine the grading, the result (or the result divided by the ULN range, depending on the test) expressed in the expected unit will be rounded to the number of decimals used for the grading.

91

<sup>\*</sup> Toxicity grading taken from FDA guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials [FDA, 2007].

<sup>\*\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

# 10.3. Appendix 3: AEs and SAEs: Definitions and procedures for recording, evaluating, follow-up, and reporting

## 10.3.1. Definition of AE

#### **AE** definition

- An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

## **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., EKG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator (i.e., not related to progression of underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New condition detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected intervention-intervention interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- Events that occur as a result of protocol-mandated procedures (i.e. invasive procedures, modification of participant's previous therapeutic regimen).

## **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments that are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital, admission for routine examination.).

- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s)
  present or detected at the start of the study that do not worsen. Pre-existing
  diseases will be recorded in the medical history section of the eCRF.
- Hospitalization for elective treatment of a pre-existing condition (known or diagnosed before signing the informed consent) that did not worsen from baseline.

## 10.3.2. Definition of SAE

An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed:

- a. Results in death
- b. Is life threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

- c. Requires inpatient hospitalization or prolongation of existing hospitalization
- In general, hospitalization signifies that the participant has been admitted (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AE. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.
- d. Results in persistent or significant disability/incapacity
- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.
- e. Is a congenital anomaly/birth defect in the offspring of a study participant
- f. Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy)
- g. Other situations:
- Possible Hy's Law case: ALT  $\geq$  3x ULN AND total bilirubin  $\geq$  2x ULN (>35% direct bilirubin) or INR >1.5 must be reported as SAE

- Medical or scientific judgment should be exercised by the investigator in deciding
  whether SAE reporting is appropriate in other situations such as significant
  medical events that may jeopardize the participant or may require medical or
  surgical intervention to prevent one of the other outcomes listed in the above
  definition. These events should usually be considered serious.
  - Examples of such events include invasive or malignant cancers, intensive treatment for allergic bronchospasm, blood dyscrasias, convulsions, or development of intervention dependency or intervention abuse.

## 10.3.3. Solicited events

## • Definition of solicited event

• Solicited events are predefined events administration site events and systemic events for which the participant is specifically questioned, and which are noted by the participant in their eDiary.

#### a. Solicited administration site events

The following administration site events will be solicited:

Table 21 Solicited administration site events

| Pain at administration site |
|----------------------------------------------------------------------|
| Redness at administration site |
| Swelling at administration site |
| Lymphadenopathy |
| (Axillary swelling/ tenderness ipsilateral to the site of injection) |

## b. Solicited systemic events

The following systemic events will be solicited:

Table 22 Solicited systemic events

| Fever |
|-------------------------|
| Headache |
| Myalgia (muscle pain) |
| Arthralgia (joint pain) |
| Fatigue (tiredness) |
| Chills |
| Abdominal pain |
| Vomiting |
| Diarrhea |

Note: Participants will be instructed to measure and record the oral temperature in the evening. If additional temperature measurements are taken at other times of the day, participants will be instructed to record the highest temperature in the eDiary.

## 10.3.4. Unsolicited AE

## **Definition of unsolicited AE**

- An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs must have been communicated by participants who signed the informed consent. Unsolicited AEs include both serious and nonserious AEs.
- Potential unsolicited AEs may be medically attended (i.e., symptoms or illnesses requiring a hospitalization, emergency room visit, or visit to/by a healthcare provider). The participants will be instructed to contact the site as soon as possible to report medically attended event(s), as well as any events that, though not medically attended, are of participant concern. Detailed information about reported unsolicited AEs will be collected by qualified site personnel and documented in the participant's records.
- Unsolicited AEs that are not medically attended nor perceived as a concern by the participant will be collected during an interview with the participants and by review of available medical records at the next visit.

# 10.3.5. Recording, assessment and follow-up of AE, SAE, AESIs and pregnancies

## 10.3.5.1. AE, SAE and AESI recording

- When an AE/SAE/AESI occurs, it is the responsibility of the investigator to review all documentation (e.g., hospital progress notes, laboratory reports, and diagnostics reports) related to the event.
- The investigator will then record all relevant AE/SAE/AESI information.
- It is not acceptable for the investigator to send photocopies of the participant's medical records to CRO in lieu of completion of the eCRF/required form.
- There may be instances when copies of medical records for certain cases are requested by CRO. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to CRO.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.
- An eDiary will be used in this study to capture solicited administration site or systemic events. The participant should be trained on how and when to complete the eDiary.
- Anyone who measures administration site or systemic events and who will record the
  event in the eDiary should be trained on using the eDiary. This training must be
  documented in the participant's source record.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

- For each solicited and unsolicited AE the participant experiences, the participant will be asked if they received medical attention (defined as unscheduled visit to or from medical personnel for any reason, including emergency room visits). This information will be recorded in the participant's eDiary (for solicited AEs) and in the participant's eCRF as part of normal AE reporting (for unsolicited AEs). If the collection of solicited AEs was not possible for any reasons via the eDiary and solicited AEs were reported to the investigator by the participant, then it would be possible for it to be reported directly to the site staff and submitted (e.g. via the eCRF). Medical attention received for SAEs/AESIs will have to be reported using the normal AE reporting process in the eCRF.
- Any unreturned eDiary will be sought from the participant through telephone call(s) or any other convenient procedure.

## 10.3.5.2. Assessment of intensity

The investigator will make an assessment of intensity for each AE, AESI and SAE reported during the study and assign it to one of the following categories:

#### • Mild:

A type of AE that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living.

## • Moderate:

A type of AE that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant.

#### • Severe:

A type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.

The intensity of the following solicited AEs will be assessed as described:

## Table 23 Intensity scales for solicited events

| Event | Intensity grade | Parameter |
|---|---|---|
| Pain at administration site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal everyday activities |
| | 2 | Moderate: Painful when limb is moved and interferes with everyday activities |
| | 3 | Severe: Significant pain at rest. Prevents normal everyday activities |
| Redness at administration site | 0 | Greatest surface diameter < 25 mm |
| | 1 | Greatest surface diameter 25 - 50 mm |
| | 2 | Greatest surface diameter 51 - 100 mm |
| | 3 | Greatest surface diameter > 100 mm |
| Swelling at administration site | 0 | Greatest surface diameter < 25 mm |
| - | 1 | Greatest surface diameter 25 - 50 mm |
| | 2 | Greatest surface diameter 51 - 100 mm |
| | 3 | Greatest surface diameter > 100 mm |
| Temperature* | 0 | < 38.0°C (100.4°F) |
| | 1 | 38.0°C (100.4°F) - 38.4°C (101.1°F) |
| | 2 | 38.5°C (101.2°F) - 38.9°C (102.0°F) |
| | 3 | >38.9°C (102.0°F) |
| Arthralgia (joint pain) | 0 | None |
| | 1 | Mild: Arthralgia present but does not interfere with activity |
| | 2 | Moderate: Arthralgia that interferes with normal activity |
| | 3 | Severe: Arthralgia that prevents normal activity |
| Headache | 0 | None |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| Fatigue (tiredness) | 0 | None |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| Lymphadenopathy | 0 | None |
| | 1 | Mild: No interference with activity |
| | 2 | Moderate: Some interference with daily activity or requires |
| | | repeated use of non-narcotic pain reliever |
| | 3 | Severe: Prevents daily activity or requires use of narcotic pain reliever |
| Chills | 0 | None |
| | 1 | Mild sensation of cold; shivering; chattering of teeth |
| | 2 | Moderate tremor of the entire body; narcotics indicated |
| | 3 | Severe or prolonged, not responsive to narcotics |
| Myalgia (muscle pain) | 0 | None |
| | 1 | Mild: Myalgia present but does not interfere with activity |
| | 2 | Moderate: Myalgia that interferes with normal activity |
| | 3 | Severe: Myalgia that prevents normal activity |
| Abdominal pain | 0 | Normal |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interferes with daily activity |
| | 3 | Severe: Prevents daily activity |

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Event | Intensity grade | Parameter |
|---|---|---|
| Vomiting | 0 | None |
| | 1 | Mild: No interference with activity or 1-2 episodes/24 hours |
| | 2 | Moderate: Some interference with activity or >2 episodes in 24 |
| | 2 | hours |
| | 2 | Severe: Prevents daily activity, requires outpatient intravenous |
| | 3 | hydration |
| Diarrhea 0 None | | None |
| | 1 | Mild: 2-3 loose stools or <400g in 24 hours |
| | 2 | Moderate: 4-5 stools or 400-800 g in 24 hours |
| | | Severe: 6 or more water stools or >800g in 24 hours |
| | 3 | or requires outpatient intravenous hydration |

<sup>\*</sup> Refer to the SoA (Section 1.3) for the definition of fever and the preferred location for temperature measurement.

## 10.3.5.3. Assessment of causality

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE/AESI. The investigator will use clinical judgment to determine the relationship.
- A *reasonable possibility* of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other
  risk factors, as well as the temporal relationship of the event to study intervention
  administration, will be considered and investigated.
- For causality assessment, the investigator will also consult the IB and/or product information, for marketed products.
- The investigator must review and provide an assessment of causality for each AE/SAE/AESI and document this in the medical notes There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to GSK. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to GSK.
- The investigator may change their opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### 10.3.5.4. Assessment of outcomes

The investigator will assess the outcome of all serious and nonserious unsolicited AEs recorded during the study as:

- Recovered/resolved
- Recovering/resolving

- Not recovered/not resolved
- Recovered with sequelae/resolved with sequelae
- Fatal (SAEs only).

## 10.3.5.5. Follow-up of AEs, SAEs, AESIs, pregnancies or any other events of interest

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by GSK to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- If a participant dies during participation in the study or during a recognized followup period, the investigator will provide GSK with a copy of any postmortem findings including histopathology.
- New or updated information will be recorded in the originally submitted documents.
- The investigator will submit any updated SAE data to GSK within 24 hours of receipt of the information.

After the initial AE/SAE/AESI/pregnancy or any other event of interest, the investigator is required to proactively follow each participant at subsequent visits/contacts. will be followed until the event is resolved, stabilized, otherwise explained, or the participant is lost to follow-up.

Other nonserious AEs be followed until the participant is lost to follow-up.

## Follow-up during the study

AEs/AESIs documented at a previous visit/contact and defined as not recovered/not resolved or recovering/resolving will be reviewed at subsequent visits/contacts until the end of the study or the participant is lost to follow-up.

If a participant dies during their participation in the study or during a recognized followup period, GSK will be provided with any available postmortem findings, including histopathology.

## Follow-up of pregnancies

Pregnant participants will be followed to determine the outcome of the pregnancy. At the end of the pregnancy, whether full-term or premature, information on the status of the mother and child will be forwarded to GSK using the electronic pregnancy report and the AE Report if applicable. Generally, the follow-up period does not need to be longer than 6 to 8 weeks after the estimated date of delivery.

Regardless of the reporting period for SAEs in this study, if the pregnancy outcome is an SAE, it should always be reported as such.

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Furthermore, the investigator must report any SAE occurring as a result of a poststudy pregnancy that is considered by the investigator to be reasonably related to the study intervention, to GSK as described in the Section 10.3.5.7.

## 10.3.5.6. Updating of SAE, AESI and pregnancy information after removal of write access to the participant's eCRF

When additional SAE, AESI or pregnancy information is received after write access to the participant's eCRF is removed, new or updated information should be recorded on the appropriate paper report, with all changes signed and dated by the investigator. The updated report should be sent to the Study contact for reporting SAEs (refer to Section 8.4.3).

## 10.3.5.7. Reporting of SAEs, AESIs and pregnancies

## SAE Reporting to CRO via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE to CRO will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) to report the event within 24 hours.
- The site will enter the SAE data into the electronic system as soon as it becomes available.
- After the study is completed at a given site, the electronic data collection tool will be taken offline to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken offline, then the site can report this information on a paper SAE form (see next section) or to the CRO by telephone.
- If the site during the course of the study or poststudy becomes aware of any serious, nonserious AEs, pregnancy exposure, related to any GSK non-IMP they will report these events to GSK or to the concerned competent authority via the national spontaneous reporting system. These will be classified as spontaneous ICSRs.
- Contacts for SAE reporting can be found in Section 8.4.7.

## SAE Reporting to CRO via Paper Data Collection Tool

- Facsimile transmission of the SAE paper data collection tool is the preferred method to transmit this information to the CRO medical monitor.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the SAE data collection tool within the designated reporting timeframes.
- Contacts for SAE reporting can be found in Section 8.4.7.

# 10.4. Appendix 4: Contraceptive guidance and collection of pregnancy information

#### 10.4.1. Definitions

#### 10.4.1.1. WOCBP

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

## 10.4.1.1.1. Women not considered as WOCBP (WONCBPs)

#### Premenarchal

Menarche is the first onset of menses in a young female. Menarche is normally preceded by several changes associated with puberty including breast development and pubic hair growth.

Additional evaluation should be considered if a participant's fertility status is unclear (e.g., amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before first dose of study intervention.

- Premenopausal female with ONE of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's: review of participant's medical records, medical examination, or medical history interview.

## Postmenopausal female

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or HRT. However, in the absence of 12 months of amenorrhea, confirmation with more than 1 FSH measurement >40 IU/L (or mIU/mL) is required.

• Females on HRT and whose menopausal status is in doubt will be required to use a non-hormonal, highly effective contraception method if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

## 10.4.2. Contraception guidance

• Female participants of childbearing potential are eligible to participate if they agree to use a highly effective contraceptive method consistently and correctly according to the methods listed in GSK's list of highly effective contraceptive methods (Table 24).

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

## Table 24 Highly effective contraceptive methods

## Highly effective contraceptive methods that are user dependenta

Failure rate of <1% per year when used consistently and correctly.

Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation

- Oral
- Intravaginal
- Transdermal

## Progestogen-only hormonal contraception associated with inhibition of ovulation

- Injectable
- Oral (if allowed by local regulation or if it is part of standard medical practice in the country).

#### Highly effective methods that are user independent

- Implantable progestogen-only hormonal contraception associated with inhibition of ovulation
- IUD
- IUS
- Bilateral tubal occlusion

#### Vasectomized partner

(A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.)

Male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant,

(The information on the male sterility can come from the site personnel's review of the participant's medical records; medical examination and/or semen analysis, or medical history interview provided by her or her partner).

#### Sexual abstinence

(Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.)

## 10.5. Appendix 5: Protocol amendment history

The Protocol Amendment Summary of Changes Table for the current amendment is located directly before the TOC.

#### Amendment 2

## **Overall Rationale for the Amendment:**

The Protocol Amendment 2 has been amended to align with the updated guidance released by the FDA on "Development and Licensure of Vaccines to Prevent COVID-19". In this guidance, the FDA indicated that safety monitoring longer than 6 months will only be "warranted for certain vaccine platforms (e.g., those that include novel adjuvants)". Hence, the follow-up of participants has been reduced from 12 months to 6 months.

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Section 1.2 (Schema), Table 1 (SoA), Table 3 (Study objectives, endpoints and estimands), Section 4.1 (Overall design), Section 4.4 (End-of-study definition), Section 8.2 (Immunogenicity assessments), Table 7 (Biological samples), Table 9 (Immunological read-outs), Section 8.4.1 (Time period and frequency for collecting AE, SAE and other safety information), Table 11 (Timeframes for collecting and reporting of safety information), Section 9.4.2.1 (Safety endpoints), Section 9.5.1 (Sequence of analyses) | Participant follow-up was reduced from 12 months to 6 months (i.e., study concludes at Visit 5 in Month 6 instead of Visit 6 in Month 12). | To align with updated FDA guidance and facilitate assessments and visits for study participants |
| LIST OF ABBREVIATIONS AND DEFINITION OF TERMS Section 10.1.3 (Informed consent process) | Deleted "Legally authorized representative" and "LAR". | "Legally authorized representative" is not applicable for this study since all participants are adults. |
| Table 1 (SoA) | Under "Unscheduled COVID-19" column, Medical History, Physical examination, Vital signs measurement, and Body temperature were added as study procedures requiring documentation in the individual eCRF. | To align with protocol text in Section 8.4.4.2.2. |
| Section 9.4.1 | Deleted "and any antipyretic taken prophylactically" | This is analysed descriptively from the Concomitant Medication eCRF. |
| Section 11 (References) | Included the reference to the guidance released by the FDA on "Development and Licensure of Vaccines to Prevent COVID-19". | This guidance serves as the basis for the amendment described above; hence, it has been included as a reference. |
| Throughout | Minor editorial and document formatting revisions. | Minor, therefore not summarized. |

## **Amendment 1**

## **Overall Rationale for the Amendment**

The Protocol Amendment 1 has been amended to comply with CBER requests, to provide clarification, to remove unnecessary restrictions, and to correct errors in the original protocol.

## **Summary of changes table of previous amendments:**

| Section # and Name | Description of Change | Brief Rationale |
|---|---|---|
| Throughout | Minor editorial and document formatting revisions | Minor; therefore, not summarized |
| Title Page | Change in Sponsor Signatory;<br>IND number was added | GSK Signatory has been changed to reflect the current Sponsor Signatory; IND number was added once available. |
| List of Abbreviations | FAS (Full Analysis Set) was removed | FAS is no longer in the protocol |
| Definition of Terms | The terms Adverse Event, Adverse Drug Reaction, Auxiliary Medicinal Product (AxMP), Background treatment, Challenge agents, Coadministered (concomitant) products, Comparator, Investigational Product, Medicinal products used to assess endpoints, Placebo, Rescue medications, Standard of Care, and SUSAR were added | These terms were added for compliance reasons |
| Section 1.1 (Synopsis), Section 1.2 (Schema); Section 4.1 (Overall design) | "multicenter" was added | To comply with a CBER request |
| Section 2.1 (Study rationale),<br>Section 5.1 (Inclusion criteria) | "the booster administered between 6 and 18 months prior to screening" was changed to "the last booster dose administered at least 6 months or more prior to screening" | To remove this unnecessary restriction in the original protocol |
| Section 2.2 (Background) | "ongoing COVID-19 pandemic" was replaced with "ongoing impact of COVID-19" | Since the pandemic is officially over |
| Table 3 (Study objectives, endpoints, and estimands) | "30" was changed to "29"; "GMTs" was changed to "GMCs"; "M6" was changed to "study conclusion"; "titers" was changed to "concentrations"; "M12" was added to the third tertiary endpoint; | To correct errors |
| Section 4.1 (Overall design) | "The study will be conducted in the United States (US)" was added | To comply with a CBER request |
| Table 4 (Study groups, intervention, and blinding) | "TC: Telephone call" was deleted from the table caption | "TC" was not present in the table |
| Section 6.3.4 (Blinding and unblinding) | "efficacy" was replaced with<br>"immunogenicity" | To correct an error |

## 219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

| Protocol Amendment 3 Final | | |
|---|---|---|
| Section # and Name | Description of Change | Brief Rationale |
| Table 15 (Analysis sets) | "Full analysis" and "Unsolicited | These are not applicable to planned |
| | safety" were deleted | analyses for this study (refer to Section 9.4 for details) |
| Table 15 (Analysis sets) | "D15 neutralizing titers against | To provide clarification |
| | pseudovirus bearing S protein from the Omicron variant of SARS-CoV- | |
| | 2" was replaced with "post-dose | |
| | specified immunogenicity data for | |
| | the relevant timepoint"; | |
| | In the Solicited Safety section, | |
| | "reported the presence or absence | |
| | of any" was added, and "safety | |
| | data" was replaced with "AE at least once" | |
| Table 15 (Analysis sets) | In the Overall Safety section, | To be consistent with planned |
| | "Unsolicited" was replaced with<br>"Exposed" | analyses |
| Section 9.4.1 (Primary endpoint) | "Exposed Set, except for solicited | To be consistent with planned |
| | AEs, which will be performed on | analyses |
| | the" was added; "and the Unsolicited Safety Set" | |
| | was deleted; | |
| Section 9.4.1 (Primary endpoint) | "screening" was replaced with "Day | To correct an error |
| , , , | 1, or if not available, closest visit | |
| | available to D1 before IMP | |
| Castian O. 4.0.0 (Insurance and initial | administration | To be a sected at with a lease of |
| Section 9.4.2.2 (Immunogenicity endpoints) | "FAS" was replaced with "Exposed Set"; | To be consistent with planned analyses |
| enapoints) | "and binding IgG Ab" was | analyses |
| | removed; | |
| | "GMCs/" was removed; | |
| | "number of doses received pre-Day | |
| | 1 and time from last dose" was | |
| Table 16 (Duate est as assisted as 5.1 | replaced with "treatment group" | This safety lab was in a discontactly. |
| Table 16 (Protocol required safety laboratory assessments) | "Prothrombin Time / INR" was added | This safety lab was inadvertently missed in this Table in the original |
| iaboratory assessificitis/ | | protocol, even though INR had been |
| | | noted in the footnote |
| Table 18 (Toxicity grading scales | "Prothrombin Time – increase by | This safety lab (i.e., Prothrombin Time) |
| for hematology parameters | factor," "1.03 – 1.10 x ULN," "1.11 | was inadvertently missed in this Table |
| evaluated in the current study) | - 1.20 x ULN," "1.21 - 1.25 x | in the original protocol |
| | ULN," and ">1.25 x ULN" were added | |
| | auueu | |

## 11. REFERENCES

Advisory Committee on Immunization Practices (ACIP). COVID-19 Vaccine Booster Dose Safety. November 19, 2021. Accessed 07 April 2023. https://www.cdc.gov/vaccines/acip/meetings/downloads/slides-2021-11-19/04-COVID-Shimabukuro-508.pdf

Centers for Disease Control (CDC). CDC COVID-19 Vaccine Task Force. Myopericarditis following COVID-19 vaccination: updates from the Vaccine Adverse Event Reporting System (VAERS). October 21, 2021. Accessed on 07 April 2023. https://stacks.cdc.gov/view/cdc/110920

Centers for Disease Control (CDC). Clinical considerations: myocarditis and pericarditis after receipt of mRNA COVID-19 vaccines among adolescents and young adults. March 23, 2023. Accessed 31 March 2023. https://www.cdc.gov/vaccines/covid-19/clinical-considerations/myocarditis.html.

European Medicines Agency (EMA). Pharmacovigilance Risk Assessment Committee (PRAC). Signal assessment report on Myocarditis, pericarditis with Tozinameran (COVID-19 mRNA vaccine (nucleoside-modified) – COMIRNATY). December 2, 2021a. Accessed 30 March 2023. https://www.ema.europa.eu/en/documents/pracrecommendation/signal-assessment-report-myocarditis-pericarditis-tozinameran-covid-19-mrna-vaccine\_en.pdf

European Medicines Agency (EMA). Pharmacovigilance Risk Assessment Committee (PRAC). Signal assessment report on myocarditis and pericarditis with Spikevax (previously COVID-19 Vaccine Moderna). December 2, 2021b. Accessed 30 March 2023. https://www.ema.europa.eu/en/documents/prac-recommendation/signal-assessment-report-myocarditis-pericarditis-spikevax-previously-covid-19-vaccine-moderna-covid\_en.pdf

Food and Drug Administration (FDA). Guidance for Industry. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. September, 2007. Accessed 07 April 2023. https://www.fda.gov/media/73679/download

Food and Drug Administration (FDA). Vaccines and Related Biological Products Advisory Committee Meeting, October 14-15, 2021. EUA amendment request for a booster dose of the Moderna COVID-19 Vaccine. October 14, 2021a. Accessed 07 April 2023. https://www.fda.gov/media/152991/download

Food and Drug Administration (FDA). Comirnaty Summary Basis for Regulatory Action (2021b). November 8, 2021b. Accessed 07 April 2023. https://www.fda.gov/media/151733/download

Food and Drug Administration (FDA). Pfizer-BioNTech COVID-19 Vaccine, Bivalent Now Authorized For All Doses. April 18, 2023a. Accessed 19 April 2023. https://www.fda.gov/emergency-preparedness-and-response/coronavirus-disease-2019-covid-19/pfizer-biontech-covid-19-vaccines

219112 (MRNA CLINRES-001) Protocol Amendment 3 Final

Food and Drug Administration (FDA). Moderna COVID-19 Vaccine, Bivalent Now Authorized For All Doses. April 18, 2023b. Accessed on 19 April 2023. https://www.fda.gov/emergency-preparedness-and-response/coronavirus-disease-2019-covid-19/moderna-covid-19-vaccines

Garcia-Beltran WF, Lam EC, St Denis K, et al. Multiple SARS-CoV-2 variants escape neutralization by vaccine-induced humoral immunity. Cell. 2021;184(9):2372-83.

Jackson LA, Anderson EJ, Rouphael NG, et al. An mRNA Vaccine against SARS-CoV-2 - Preliminary Report. N Engl J Med. 2020;383(20):1920-1931.

Mathieu E, Ritchie H, Rodés-Guirao L, et al. Coronavirus Pandemic (COVID-19). March 03, 2023. Accessed on 23 March 2023. https://ourworldindata.org/coronavirus

Peeples, L. News Feature: Avoiding pitfalls in the pursuit of a COVID-19 vaccine. Proc Natl Acad Sci USA. 2020;117(15): 8218-21.

Rüggeberg JU, Gold MS, Bayas JM, et al. Anaphylaxis: case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2007;25(31):5675-84.

Sexson Tejtel SK, Munoz FM, Al-Ammouri I, et al. Myocarditis and pericarditis: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2022;40(10):1499-511.

World Health Organization [WHO]. Advice for the public: Coronavirus disease (COVID-19). March 18, 2023. Accessed 31 March 2023. https://www.who.int/emergencies/diseases/novel-coronavirus-2019/advice-for-public

Zhou B, Thao TTN, Hoffmann D, et al. SARS-CoV-2 spike D614G change enhances replication and transmission. Nature. 2021;592(7852):122-7.

## Signature Page for 219112 TMF-18266190 v1.0

| Reason for signing: Approved | Name: PPD |
|---|---|
| | Role: Approver |
| | Date of signature: 07-Feb-2024 13:11:36 GMT+0000 |

Signature Page for TMF-18266190 v1.0